

# Statistical Analysis Plan

Protocol Number: AX-158-101

A Randomised, Double-blind, Placebo-controlled, Study of the Safety,
Tolerability, and Pharmacokinetics of AX-158 Following
Administration of Single and Multiple Ascending Oral Doses and Food
Effect sub-study in Healthy Male Volunteers

Simbec-Orion Protocol ID: RD 675/34625

Prepared for: **Artax Biopharma Inc.** 

Prepared by:

Simbec-Orion Clinical Pharmacology

Unit 29 Merthyr Industrial Park,

Merthyr Tydfil CF48 4DR

Tel: +44 (0) 1443 690977

CONFIDENTIAL

**Version** Final 1.0

**Author** Alexandra Soós



# Statistical Analysis Plan

Protocol Number: AX-158-101

A Randomised, Double-blind, Placebo-controlled, Study of the Safety,
Tolerability, and Pharmacokinetics of AX-158 Following
Administration of Single and Multiple Ascending Oral Doses and Food
Effect sub-study in Healthy Male Volunteers

Simbec-Orion Protocol ID: RD 675/34625

| Author: | Alexandra | Soós |
|---------|-----------|------|

Version: Final I.0

The undersigned have reviewed and revised this SAP and find it to be consistent with the study requirements:

| DocuSigned by: | |
|---|---|
| Kerry Williams | |
| Signer Name: Kerry Williams Signing Reason: I have reviewed this document Signing Time: 14-Dec-2022 17:36 GMT | |
| F3E94C122FE94BD1802DA6C1E65CE70F | |
| Kerry Williams, Statistics Team Lead, Simbec-Orion Clinical Pharmacology | Date |
| DocuSigned by: | |
| Gennifer Derham | |
| Signer Name: Jennifer Derham Signing Reason: I approve this document Signing Time: 14-Dec-2022 17:35 GMT | |
| 0A4B17FF670748EFAEEFF9C32466E9C1 | |
| Jennifer Derham, Project Manager, Simbec-Orion Clinical Pharmacology | Date |

Version: 3.0

Document Title: SA

Document Title:SAP Template - Phase 1Document Number:TEMP-00109Previous Document Number:STATt008



# Artax Biopharma Inc: AX-158-101 Statistical Analysis Plan Final v1.0 14DEC2022

| DocuSigned by: Signer Name: Simon Hutchings Signing Reason: I approve this document Signing Time: 15-Dec-2022 08:56 GMT E123B8AADABB4493AD2B860956A17BB0 | |
|---|---|
| Simon Hutchings, Director of Pharmacology, Simbec-Orion Clinical | Date |
| Pharmacology | |
| DocuSigned by: Sult Batty Signer Name: Scott Batty Signing Reason: I approve this document Signing Time: 15-Dec-2022 09:28 EST DC9E14FC9DC84708AD921E2E6124D8E4 | Date |
| Dr. Scott Batty, MD, Chief Medical Officer, Artax Biopharma | Date |

Version:
Document Title:
Document Number:
Previous Document Number:

3.0 SAP Template - Phase 1 TEMP-00109 STATt008



# TABLE OF CONTENTS

| I | INTRU | JDUCTION | δ |
|----|-------|-------------------------------------------|----|
| | 1.1 | GENERAL | 8 |
| | 1.2 | CHANGES FROM PROTOCOL | 8 |
| | 1.3 | CHANGES FROM PREVIOUS VERSIONS OF THE SAP | 8 |
| 2 | STUD | Y OBJECTIVES | 8 |
| 3 | STUD | Y DESIGN | 8 |
| | 3.1 | OVERVIEW | 9 |
| | 3.2 | INCLUSION AND EXCLUSION CRITERIA | 10 |
| | 3.3 | STUDY TREATMENT | 10 |
| | 3.4 | STUDY TIMEPOINTS | 11 |
| | 3.4.1 | Schedule of Study Procedures | 11 |
| | 3.5 | SAMPLE SIZE CONSIDERATIONS | 13 |
| | 3.6 | RANDOMISATION | 14 |
| 4 | STUD | Y VARIABLES AND COVARIATES | 14 |
| | 4.1 | PRIMARY VARIABLES | 14 |
| | 4.2 | SECONDARY VARIABLES | 14 |
| 5 | DEFIN | IITIONS AND DERIVED VARIABLES | |
| 6 | ANAL | YSIS SETS | |
| | 6.1 | ALL CONSENTED SET | 16 |
| | 6.2 | SAFETY SET | 16 |
| | 6.3 | PK SET | 16 |
| 7 | SAFET | TY MONITORING | 17 |
| 8 | INTER | IM ANALYSES | 17 |
| 9 | DATA | | 17 |
| | 9.1 | eCRF Data | |
| | | EXTERNAL DATA | |
| | 9.2.1 | Laboratory Data | |
| | 9.2.2 | Other non-CRF data | |
| | 9.3 | RANDOMISATION LIST | 19 |
| | 9.4 | PROGRAMMING AND DATA REVIEW | 19 |
| 10 | STATI | STICAL METHODS | 19 |
| | 10.1 | GENERAL PRINCIPLES | 19 |
| | 10.2 | STRATIFICATION AND COVARIATE ADJUSTMENT | 20 |
| | 10.3 | INTERACTIONS | |
| | 10.4 | MISSING DATA | 20 |

Version:

Document Title: SAP Template - Phase 1
Document Number: TEMP-00109
Previous Document Number: STATt008





| | 10.5 | POOLING OF SITES | 21 |
|----|--------|------------------------------------------|-----|
| | 10.6 | Multiple Comparisons | 21 |
| | 10.7 | SUBGROUP ANALYSES | 21 |
| | 10.8 | STATISTICAL ISSUES | 21 |
| 11 | STATIS | STICAL OUTPUT | 21 |
| | 11.1 | SUBJECT DISPOSITION | 21 |
| | 11.2 | SUBJECT CHARACTERISTICS AT BASELINE | 22 |
| | 11.2.1 | Demographic and Baseline Characteristics | 22 |
| | 11.3 | EFFICACY ANALYSES | 22 |
| | 11.4 | PK ANALYSES | 22 |
| | 11.4.1 | Concentration Data | 22 |
| | 11.4.2 | Derived PK Parameters | 23 |
| | 11.4.3 | Statistical Analysis of PK Data | 31 |
| | 11.5 | PD ANALYSES | 34 |
| | 11.6 | SAFETY ANALYSES | 34 |
| | 11.6.1 | Adverse Events | 34 |
| | 11.6.2 | Laboratory Data | 35 |
| | 11.6.3 | Vital Signs | 36 |
| | 11.6.4 | Electrocardiogram | 36 |
| | 11.7 | OTHER | 37 |
| | 11.7.1 | Prior and Concomitant Medication | 37 |
| | 11.7.2 | All Other Data | 38 |
| 12 | VALID | ATION | 38 |
| 13 | LITERA | ATURE CITATIONS/REFERENCES | 38 |
| 14 | LIST O | F TABLES, FIGURES AND LISTINGS | 39 |
| 15 | SHELL | S FOR TABLES, FIGURES AND LISTINGS | 44 |
| 16 | APPEN | DICES | 106 |
| | 16.1 | Normal Ranges | 106 |



# **GLOSSARY OF ABBREVIATIONS**

| ADaM | Analysis Data Model |
|---|---|
| AE | Adverse Event |
| ANCOVA | Analysis of Covariance |
| ANOVA | Analysis of Variance |
| ATC | Anatomical Therapeutic Chemical |
| AUC | Area Under the Concentration Curve |
| AUC <sub>%extrapolated</sub> | Residual Area |
| AUC <sub>0-inf</sub> | Area Under the Concentration-time Curve calculated from the time of |
| ACC0-inf | dosing to infinity |
| AUC <sub>0-r</sub> | Area Under the Concentration-time Curve calculated from the time of |
| 710 00-1 | dosing to the last measurable concentration |
| AUC <sub>0-tau</sub> | Area Under the Concentration-time Curve calculated over one dosing |
| | interval at steady state |
| BLQ | Below Limit of Quantification |
| BMI | Body Mass Index |
| CDISC | Clinical Data Interchange Standards Consortium |
| CI | Confidence Interval |
| CL | Total body clearance |
| CL <sub>ss</sub> | Total body clearance at steady state |
| C <sub>max</sub> | Maximum observed concentration |
| C <sub>min</sub><br>CRA | Minimum observed concentration |
| CRF | Clinical Research Associate |
| CRO | Case Report Form Clinical Research Organisation |
| CS | Clinically Significant |
| CSR | Clinical Study Report |
| CV | Coefficient of Variation |
| DBL | Database Lock |
| DMP | Data Management Plan |
| DOB | Date of Birth |
| DRM | Data Review Meeting |
| ECG | Electrocardiogram |
| eTMF | Electronic Trial Master File |
| GM | Geometric Mean |
| h | Hours |
| ICH | International Conference on Harmonisation |
| IMP | Investigational Medicinal Product |
| $K_{el}$ | Elimination rate constant |
| LLOQ | Lower Limit of Quantification |
| LSMean | Least Squares Mean |
| MedDRA | Medical Dictionary for Regulatory Activities |
| mg | Milligram |
| ml | Millilitre |
| N | Number of subjects in the analysis set |
| n | Number of subjects with non-missing observations |
| NCS | Not clinically significant |
| PD | Pharmacodynamics |


**Document Title:** SAP Template - Phase 1

Document Number: TEMP-00109
Previous Document Number: STATt008



# Artax Biopharma Inc: AX-158-101 Statistical Analysis Plan Final v1.0 14DEC2022

| PK | Pharmacokinetics |
|------------------|--------------------------------------------------------|
| PT | Preferred Term |
| QC | Quality Control |
| SAE | Serious Adverse Event |
| SAP | Statistical Analysis Plan |
| SD | Standard Deviation |
| SDTM | Study Data Tabulation Model |
| SE | Standard Error |
| SOC | System Organ Class |
| t <sub>1/2</sub> | Terminal phase half life |
| TEAE | Treatment Emergent Adverse Event |
| TFL | Tables, Figures and Listings |
| $T_{max}$ | Time from dosing to the maximum observed concentration |
| TMF | Trial Master File |
| Vz | Apparent volume of distribution |
| WHO | World Health Organisation |
| WHODD | World Health Organisation Drug Dictionary |
| μg | Microgram |


Document Title: SAP Template - Phase 1
Document Number: TEMP-00109
Previous Document Number: STATt008



# 1 INTRODUCTION

#### 1.1 GENERAL

This statistical analysis plan (SAP) describes the statistical methods to be used during the reporting and analyses of data collected under the AX-158-101 protocol dated 15 March 2022 and should be read in conjunction with the study protocol and electronic case report form (eCRF).

This version of the plan has been developed using protocol version 5.0 dated 15 March 2022 and annotated CRF version 4.3 dated 22AUG2022 further changes to the protocol or eCRF will be reviewed for potential impact on the SAP which will be amended if it is deemed necessary.

Draft versions of the SAP will undergo review by the Statistical Reviewer, Statistical Programmer, Project Manager, PK Analyst, Medical Writer, Principal Investigator and the Sponsor/Sponsor representative. The analysis plan will be finalised and approved by the Sponsor prior to Database Lock (DBL).

### 1.2 CHANGES FROM PROTOCOL

The PK Set criterion of having at least one PK sample with concentration above the lower limit of quantitation (LLOQ) has been removed to enable inclusion of subjects with all-BLQ profiles to contribute to the concentration data summaries.

For Part B the statistical analysis (ANOVA) will be performed including fixed effects for sequence, period, treatment and subject nested within sequence.

# 1.3 CHANGES FROM PREVIOUS VERSIONS OF THE SAP

Not applicable.

# 2 STUDY OBJECTIVES

### Primary Objective(s):

• To assess the safety and tolerability of single and multiple ascending doses of AX-158 when administered to healthy participants (Part A and Part C)

### **Secondary Objective(s):**

- To investigate the PK of single and multiple doses of AX-158 in healthy participants (Part A and Part C).
- To investigate any food effect on the PK of AX-158 following oral administration of a single dose to healthy participants (Part B).

# 3 STUDY DESIGN





#### 3.1 OVERVIEW

This is a phase I, randomised, double-blind, placebo-controlled study to investigate the safety, tolerability, and PK of AX-I58 in healthy male participants following single (Part A) and multiple (Part C) ascending doses including food effect (Part B).

The study will be conducted in three parts:

#### Part A

Part A (SAD) will enrol up to 8 participants per cohort randomised (3:1) to receive AX-158 or placebo. Part A will follow a single ascending dose (SAD) design with all participants receiving one dose of AX-158 (or placebo) in the fasted state.

This part will be conducted in up to 34 participants (8 participants in cohorts I and 5, 6 participants in cohorts 2, 3 and 4). An additional two cohorts of up to eight (8) participants each (up to 16 additional participants total) may be investigated if required.

## Part B

Part B (Food Effect) will be conducted in up to 8 participants in a cross-over manner; each participant will receive AX-158 in the fed and fasted state.

This part will be conducted in up to 8 participants in a cross-over manner.

### Part C

Part C (MAD) will enrol up to 8 participants per cohort randomised to (3:1) to receive AX-158 or placebo. Part C will follow a multiple ascending dose (MAD) design with participants receiving AX-158 (or placebo) once daily for 10 consecutive days, in a fed or fasted state (depending on the outcome of the Part B (Food Effect). Doses, dosing duration and dose regimen (i.e., q.i.d., b.i.d., t.i.d.) of AX-158 and matching placebo for Part C may be modified based on all available safety, tolerability, and PK data and applied to additional MAD cohorts.

This part will be conducted in up to twenty-four (24) participants (3 cohorts of up to 8 participants). An additional two cohorts of up to eight (8) participants each (up to 16 additional participants total) may be investigated if required.

Duration of study:

- Part A: approximately 6 weeks for each individual (from the screening to post-study follow-up).
- Part B: approximately 8 weeks for each individual (from the screening to post-study follow-up).
- Part C: approximately 7 weeks for each individual (from the screening to post-study follow-up).

A review of safety data and available preliminary PK data will be conducted by the DERC (Dose Escalation Review Committee). Following DERC review of data from Part A, the dose for participants in Part B will be determined. Following DERC review of data from Part B, the dose for participants in Part C will be determined, and cohorts in Part C may be administered AX-158 under fasted or fed conditions as deemed appropriate, pending DERC determination of any appreciable impact of food on the absorption, distribution, metabolism, and excretion (ADME) of AX-158.



# 3.2 INCLUSION AND EXCLUSION CRITERIA

To be eligible for inclusion into this study, each subject must fulfil all inclusion criteria and not violate any exclusion criteria (for the protocol under which they are entered) during screening prior to randomisation. Details of the inclusion and exclusion criteria are presented within the protocol (section 10.5).

### 3.3 STUDY TREATMENT

For <u>Part A (SAD)</u>, 5 planned cohorts of 8 subjects (with an option to include up to 2 additional cohorts) will receive the following in accordance with the randomisation schedule:

- a single dose of AX-158 capsules (6 subjects)
- matching placebo (2 subjects)

The IMPs will be administered fasted with 240 ml water.

For Part B (Food Effect), I cohort of 8 subjects will receive a single dose of AX-158 capsules in either the fed or fasted state over 2 periods (I per period) in accordance with the randomisation schedule.

For <u>Part C (MAD)</u>, 3 cohorts of 8 subjects (with an option to include up to 2 additional cohorts) will receive the following in accordance with the randomisation schedule:

- AX-158 capsules for 10 days (6 subjects)
- matching placebo for 10 days (2 subjects)

The IMPs will be administered fasted with 240 ml water.

If a food effect is observed in Part B, cohorts in Part C may be dosed with a standardised meal.

For Part A (SAD) and Part C (MAD), a dose leader design will be implemented with 2 participants being dosed on the first dosing day of each cohort. Of these 2, I will be on active drug and I on placebo.



#### 3.4 STUDY TIMEPOINTS

# 3.4.1 Schedule of Study Procedures

#### Part A

| Visits <sup>1,2</sup> | | Treatment Period | | | | | | | | | | | | Follow up | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visits <sup>1,2</sup> | Screening | | In-house | | | | | | | | | | | | | | | |
| Days | Day - 28<br>to -2 | Day<br>- 1 | Day 1 Post- Post- Treatment Treatment Treatment 1 (Day 2) 2 (Day 3) 3 (Day 4) | | | | | | | | | Treatment | 5-7 days from<br>last IMP dose | | | | | |
| Time (h) | | | Pre-<br>Dose | 0 | 0.5 | 0.75 | 1h | 2h | 3h | 4h | 6h | 8h | 12h | 24h | 36h | 48h | 72h | |
| Informed Consent | X | | | | | | | | | | | | | | | | | |
| Inclusion/Exclusion3 | X | X | X | | | | | | | | | | | | | | | |
| Demographics | X | | | | | | | | | | | | | | | | | |
| Height/Weight/BMI | X | X | | | | | | | | | | | | | | | | |
| Medical History &<br>Concurrent<br>Conditions | x | | | | | | | | | | | | | | | | | |
| Virology Tests<br>(HIV, HBsAg,<br>HCV) | х | | | | | | | | | | | | | | | | | |
| Drug and Alcohol<br>Screen <sup>5</sup> | Х | х | | | | | | | | | | | | | | | | |
| COVID-19 Test | | X | | | | | | | | | | | | | | | | |
| Biochemistry | $X^6$ | X | | | | | | | | | | | | X | | | X | X |
| Haematology | X | X | | | | | | | | | | | | X | | | X | X |
| Urinalysis | X | X | | | | | | | | | | | X | X | | | X | X |
| Coagulation <sup>7</sup> | X | X | | | | | | | | | | | | X | | | X | X |
| Randomisation | | | X | | | | | | | | | | | | | | | |
| Adverse Events | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Vital Signs <sup>8</sup> | X | X | X | | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Physical<br>Examination | x | $X^{11}$ | | | | | | | | | | | | | | | X <sup>11</sup> | X <sup>11</sup> |
| 12-Lead ECG9 | X | X | X | | X | | | | | X | | | X | X | | X | X | X |
| Prior & | | | | | | | | | | $\overline{}$ | $\overline{}$ | | | | | | | |
| Concomitant<br>Medication | X | X | X | X | X | X | X | X | X | х | Х | Х | X | X | X | x | X | X |
| Dose IMP <sup>10</sup> | | | | X | | | | | | | | | | | | | | |
| Blood Sampling for<br>PK | | | X | | Х | х | Х | X | X | х | Х | X | Х | х | х | x | x | |
| Exploratory PD sample | | | X <sup>12</sup> | | | | | | | | | | | | | | | |

- I. All cohorts will complete only I Treatment Period.
- 2. Participants will be in the clinical unit for their in-house period from the morning before dosing (Day -1), until the completion of all the assessments on Post-Treatment 3 (Day 4).
- 3. Eligibility will be determined during screening. Continued eligibility will be confirmed on Day -1, and pre-dose Day 1.
- 4. Height measured at Screening only.
- 5. A urine sample will be used to screen for drugs of abuse (including alcohol and cotinine).
- 6. Total serum testosterone only required at screening.
- 7. Coagulation testing INR, aPTT and PT.
- 8. Vital signs include the following assessments: supine systolic and diastolic blood pressure, supine heart rate, respiration rate and oral temperature
- 9. 12-lead ECG will be performed at screening, each period pre-dose and at 30 min, 4 h, 12 h, 24 h, 48 h and 72 h post-dose and at the post-study follow up visit.
- 10. IMP or placebo will be administered orally in a fasted state (after an overnight fast of at least 10 h) with 240 mL water. The fast will be broken 4 h post-dose with lunch.
- 11. Symptom directed
- 12. Cohort 3 onwards additional samples will be taken based on emerging data



#### Part B

| Visits <sup>1,2</sup> | Screening | | Treatment Periods 1 & 2 | | | | | | | | | | | | Follow up | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visits | Screening | | In-house | | | | | | | | | | | ronow up | | | | |
| Days | Day - 28<br>to -2 | Day<br>- 1 | | Day 1 Post- Post- Treatment Treatment 1 (Day 2) 2 (Day 3) 3 (Day 4) | | | | | | | | | 5-7 days from last<br>IMP dose | | | | | |
| Time (h) | | | Pre-<br>Dose | 0 | 0.5 | 0.75 | 1h | 2h | 3h | 4h | 6h | 8h | 12h | 24h | 36h | 48h | 72h | |
| Informed Consent | X | | | | | | | | | | | | | | | | | |
| Inclusion/Exclusion3 | X | X | X | | | | | | | | | | | | | | | |
| Demographics | X | | | | | | | | | | | | | | | | | |
| Height/Weight/BMI4 | X | X | | | | | | | | | | | | | | | | |
| Medical History &<br>Concurrent<br>Conditions | x | | | | | | | | | | | | | | | | | |
| Virology Tests<br>(HIV, HBsAg,<br>HCV) | х | | | | | | | | | | | | | | | | | |
| Drug and Alcohol<br>Screen <sup>5</sup> | X | X | | | | | | | | | | | | | | | | |
| COVID-19 Test | | X | | | | | | | | | | | | | | | | |
| Biochemistry | X <sup>6</sup> | X | $X^6$ | | | | | | | | | | | X | | | X | X |
| Haematology | X | X | | | | | | | | | | | | X | | | X | X |
| Urinalysis | X | X | | | | | | | | | | | X | X | | | X | X |
| Coagulation <sup>7</sup> | X | X | | | | | | | | | | | | X | | | X | X |
| Randomisation | | | X | | | | | | | | | | | | | | | |
| Adverse Events | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Vital Signs <sup>8</sup> | X | X | X | | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Physical<br>Examination | X | X <sup>11</sup> | | | | | | | | | | | | | | | X <sup>11</sup> | X <sup>11</sup> |
| 12-Lead ECG9 | X | X | X | | X | | | | | X | | | X | X | | X | X | X |
| Prior & Concomitant<br>Medication | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | Х |
| Dose IMP <sup>10</sup> | | | | X | | | | | | | | | | | | | | |
| Blood Sampling for<br>PK | | | X | | X | X | X | X | X | X | Х | X | X | X | X | X | X | |

- I. All cohorts will complete Treatment Period I & 2.
- 2. For Treatment Periods I & 2, participants will be in the clinical unit for their in-house period from the morning before dosing (Day -I), until the completion of all the assessments on Post-Treatment 3 (Day 4).

  3. Eligibility will be determined during screening. Continued eligibility will be confirmed on Day -I, and pre-dose Day I for Treatment Periods I & 2.
- 4. Height measured at Screening only.
- 5. A urine sample will be used to screen for drugs of abuse (including alcohol and cotinine). 6. Total serum testosterone required at screening and pre-dose DI each treatment period (Biochemistry sample: pre-dose Day I total serum testosterone only).
- 7. Coagulation testing INR, Aptt and PT.
- 8. Vital signs include the following assessments: supine systolic and diastolic blood pressure, supine heart rate, respiration rate and oral temperature
- 9. 12-lead ECG will be performed at screening, each period pre-dose and at 30 min, 4 h, 12 h, 24 h, 48 h and 72 h post-dose and at the post-study follow up visit.
- 10. Participants will receive a single dose of AX-158 following an overnight fast of at least 10 h OR following consumption of a high-fat breakfast over 2 treatment periods (I per period). AX-158 should be administered 30 mins after the start of the meal. II. Symptom directed



#### Part C

| Visits <sup>1</sup> | Screening | | In-house | | | | | | | | | | | | | Follow<br>up | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Days | Day - 28<br>to -2 | Day – 1 | | Day 1-4, Day 10-13 <sup>15</sup> | | | | | | | | | Day 5-9 | 5-7<br>days<br>from<br>last<br>IMP<br>dose | | | | | |
| Time (h) | | | Pre-<br>Dose | 0 | 0.5 | 0.75 | 1h | 2h | 3h | 4h | 6h | 8h | 12h | 24h | 36h | 48h | 72h | | |
| Informed Consent | X | | | | | | | | | | | | | | | | | | |
| Inclusion/Exclusion <sup>2</sup> | X | X | X | | | | | | | | | | | | | | | | |
| Demographics | X | | | | | | | | | | | | | | | | | | |
| Height/Weight/BMI3 | X | X | | | | | | | | | | | | | | | | | |
| Medical History &<br>Concurrent Conditions | X | | | | | | | | | | | | | | | | | | |
| Virology Tests (HIV,<br>HbsAg, HCV) | X | | | | | | | | | | | | | | | | | | |
| Drug and Alcohol<br>Screen <sup>4</sup> | X | X | | | | | | | | | | | | | | | | | |
| COVID-19 Test | | X | | | | | | | | | | | | | | | | $X^{15}$ | |
| Biochemistry | $X^7$ | X | $X^{7,8}$ | | | | | | | | | | | $X^{7,8}$ | | | X | X <sup>6,7,8</sup> | X |
| Haematology | X | X | | | | | | | | | | | | X | | | X | $X^6$ | X |
| Urinalysis | X | X | | | | | | | | | | | X | X | | | X | X <sup>6</sup> | X |
| Coagulation <sup>5</sup> | X | X | | | | | | | | | | | | X | | | X | $X^6$ | X |
| Randomisation | | | X | | | | | | | | | | | | | | | | |
| Adverse Events | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Vital Signs <sup>9</sup> | X | X | X | | X | X | X | X | X | X | X | X | X | X | X | X | X | X <sup>6</sup> | X |
| Physical Examination | X | $X^{13}$ | | | | | | | | | | | | | | | $X^{13}$ | | $X^{13}$ |
| 12-Lead ECG <sup>10</sup> | X | X | X | | X | | | | | Х | | | X | X | | X | X | X <sup>6</sup> | X |
| Prior and Concomitant<br>Medication | Х | X | х | x | х | Х | х | x | х | х | х | х | х | Х | Х | х | Х | X | х |
| Dose IMP <sup>11</sup> | | | | Х | | | | | | | | | | X | | X | X | X | |
| Blood Sampling for PK | | | X | | X | X | Х | X | Х | Х | Х | Х | X | X | Х | X | X | X14 | |
| Urine Sampling for PK Exploratory PD sample | | | X <sup>12</sup> X <sup>16</sup> | 4 | | | | | | | | | | | | | | | |

- 1. For each cohort participants will be in the clinical unit for their inpatient visit from the morning before dosing (Day -1), until the completion of all assessments on Day 13.
- 2. Eligibility will be determined during screening. Continued eligibility will be confirmed on Day -1, and pre-dose Day 1-10
- 3. Height measured at Screening only.
- 4. A urine sample will be used to screen for drugs of abuse (including alcohol and cotinine)
- 5. Coagulation testing INR, aPTT and PT
- 6. Pre dose on Day 5 only
- 7. Total serum testosterone required at screening, fasted pre dose D1, D5 and on D11 (Biochemistry sample: pre-dose Day1 total serum testosterone only)
- 8. Serum LH required at pre-dose DI, D5 and on DII (Biochemistry sample: pre-dose DayI serum LH only)
- 9. Vital signs include the following assessments: supine systolic and diastolic blood pressure, supine heart rate, respiration rate and oral temperature
- 10. 12-lead ECG will be performed at screening, pre-dose and at 30 min, 4 h, 12 h, 24 h, 48 h and 72 h post-dose Days I and 10 and at the post-study follow up visit.
- II. For all cohorts IMP or placebo will be administered orally in a fasted state (after an overnight fast of at least 10 h) with 240 mL water. The fast will be broken 4 h post-dose with lunch on Days 1-10.
- 12. Urine sampling: for AX-158: pre-dose and in intervals of 0-12, 12-24, 24-48 and 48-72 h post-dose on Day 1 and Day 10
- 13. Symptom Directed
- 14. Pre-dose trough sample day 5 only
- 15. COVID-19 test on day 8 and prior to check out.
- 16. Additional samples will be taken based on emerging data

#### 3.5 SAMPLE SIZE CONSIDERATIONS

The sample size chosen for this study is not based on a formal statistical estimation but is considered adequate to meet the objectives of the study. A sufficient number of participants will be initially screened for enrolment to ensure that the planned sample size is achieved.


**Document Title:** SAP Template - Phase 1

Document Number:TEMP-00109Previous Document Number:STATt008



#### 3.6 RANDOMISATION

Simbec-Orion using the PROC PLAN procedure of SAS® (9.4 or higher or EG). The randomisation code will include 2 dose-leaders (1 active:1 placebo) in each cohort (for Part A and Part C only).

#### Part A

Format and range of randomisation numbers: 101 - 156. Replacement subjects will be assigned the same randomisation as the participant they are replacing, however, 300 will be added to the number (i.e., 401 would replace 101 etc.).

The following IMPs will be used: AX-158 capsules vs Placebo.

#### Part B

Format and range of randomisation numbers: 201 - 208. Replacement subjects will be assigned the same randomisation as the participant they are replacing, however, 300 will be added to the number (i.e., 501 would replace 201 etc.).

The following IMPs will be used: AX-158 capsules in fed/fasted state.

| Sequence | Period I | Period 2 |
|----------|-----------------|-----------------|
| 1 | AX-158 - Fasted | AX-158 - Fed |
| 2 | AX-158 - Fed | AX-158 - Fasted |

#### Part C

Format and range of randomisation numbers: 301 - 340. Replacement subjects will be assigned the same randomisation as the participant they are replacing, however, 300 will be added to the number (i.e., 601 would replace 301 etc.).

The following IMPs will be used: AX-158 capsules vs Placebo.

# 4 STUDY VARIABLES AND COVARIATES

#### 4.1 PRIMARY VARIABLES

The primary safety endpoints for this study are as follows:

- Adverse events
- Laboratory safety parameters (biochemistry, hematology, coagulation, urinalysis)
- Vital signs (systolic/diastolic blood pressure, heart rate, oral body temperature and respiratory rate)
- 12-Lead ECG (Heart rate, PR interval, QRS width, RR interval, QT interval and QT interval corrected using Fredericia's formula (QTcF)

#### 4.2 SECONDARY VARIABLES

The secondary plasma pharmacokinetic (PK) endpoints for this study are as follows:

C<sub>max</sub> Maximum observed concentration

Version: 3.0 Document Title: SA

 Document Title:
 SAP Template - Phase 1

 Document Number:
 TEMP-00109

 Previous Document Number:
 STATt008





T<sub>max</sub> Time to maximum observed concentration
 T<sub>lag</sub> The delay in achieving T<sub>max</sub> (only in Part B)

 $\begin{array}{ll} \bullet & k_{el} & & \text{Elimination rate constant} \\ \bullet & t_{1/2} & & \text{Terminal elimination half-life} \end{array}$ 

ullet AUC<sub>0-24</sub> Area under the concentration-time curve (AUC) from the time of dosing

to 24 hour post dose

• AUC<sub>0-tau</sub> If part C dosing is not q.d.

AUC<sub>0-t</sub>
 Area under the concentration-time curve (AUC) from the time of dosing

to the time of the last measurable concentration

AUC<sub>0-inf</sub>
 AUC extrapolated to infinity

 $\bullet \quad \mathsf{AUC}_{\text{$^{\texttt{extrapolated}}}} \qquad \quad \mathsf{Residual} \; \mathsf{area}$ 

CL/F Apparent total body clearance
 Vz/F Apparent volume of distribution

The secondary urine PK endpoints for Part C of this study are:

Ae
 Amount and cumulative amount of dose excreted in urine over each

collection interval

Ae% % and cumulative % of dose excreted in urine over each collection interval

• CL<sub>R</sub> Renal clearance

# 5 DEFINITIONS AND DERIVED VARIABLES

**Treatment/IMP:** Treatment or IMP is taken to mean either AX-158 at all dose levels, in the fed or fasted state, or placebo.

**Baseline:** For Part A and Part C unless stated otherwise, baseline is defined by subject and by variable as the last non-missing value (including repeat/unscheduled assessments) before the first dose of study drug.

For Part B unless stated otherwise, baseline is defined by subject and by variable as the last non-missing value (including repeat/unscheduled assessments) before the first dose of study drug in each treatment period. This will normally be the pre-dose assessment on Day I of each treatment period but if this assessment is missing (or not planned) then the last assessment prior to first dose in Period I will be used instead, if available. Specific baselines for each endpoint are defined in Section II, where appropriate.

**Study Day**: Study day is the number of days since start of treatment where the date of first dose is counted as Day I.

**Blood Sampling Time Deviation:** Actual sample time – planned sample time.

**Protocol Deviation:** a deviation related to study inclusion or exclusion criteria, conduct of the trial, subject management or subject assessment. This refers to any change, divergence, or departure from the study design or procedures defined in the protocol. Protocol deviations captured in the CRF will be discussed at the Data Review Meeting (DRM) before Database Lock (DBL). In addition, any deviations


**Document Title:**SAP Template - Phase 1 **Document Number:**TEMP-00109

Previous Document Number: STA

STATt008





identified during the DRM will be discussed and included in the database as necessary. All protocol deviations within the study database will be classified as either 'Major' or 'Minor' prior to DBL, details of which will be included within the Protocol Deviations listing.

# 6 ANALYSIS SETS

Membership of the analysis sets will be reviewed during the DRM and agreed prior to DBL. These will be reviewed by the Sponsor, Study Statistician, PK Analyst and Project Manager and included within the DRM minutes. Where PK data is not available at the time of DBL, subjects will be assumed to be included in the analysis set unless the PK data provide reason to exclude a subject, in which case this will be discussed with the Sponsor and documented within the Analysis Sets listing (Listing 16.2.3.1).

#### 6.1 ALL CONSENTED SET

All subjects for whom informed consent was obtained will constitute the All Consented Set.

This analysis set will be used for the study disposition listing and summary.

#### 6.2 SAFETY SET

All randomised subjects who receive at least 1 dose of IMP will be included in the Safety Set.

This analysis set will be used for baseline and safety summaries as well as for all study listings.

# 6.3 PK SET

The PK set will include subjects who receive active IMP (one dose in Part A, both doses in Part B (fed/fasted), up to 10 doses in Part C), have sufficient plasma concentration-time profiles and comply with the following criteria:

- Do not have an occurrence of vomiting (that occurs at or before 2 times median T<sub>max</sub> within the appropriate cohort or treatment) or diarrhoea which renders the concentration profile unreliable. For Part C this applies to PK sampling days only.
- Do not use a concomitant medication which renders the concentration profile unreliable.
- Do not have a Day I pre-dose concentration that is greater than 5% of the corresponding C<sub>max</sub>.
- Do not violate the protocol in such a way that may invalidate or bias the results (major protocol violators).

For Part C, a subject may be included in the PK Set if they have a valid Day I PK profile which meets the above criteria, as the Day I PK data can be included in the dose proportionality/independence assessment. For inclusion in the Day I0 dose proportionality/independence assessment, subjects must have fulfilled the above criteria and received all doses of study drug.

In order to be included in the statistical comparisons for Part B, a subject is required to be included in the PK Set for the two treatments being evaluated within the particular comparison.

All protocol deviations within the study database will be reviewed to determine whether they affect a subject's eligibility for inclusion in the PK Set. Any deviations and reasons for exclusion will be identified and documented before statistical analysis of the pharmacokinetic data is undertaken.

Version:
Document Title:
Document Number:
Previous Document Number:

SAP Template - Phase 1 TEMP-00109 STATt008



This analysis set will be used for PK summaries and statistical analyses.

# 7 SAFETY MONITORING

Following completion of each cohort, a summary of all relevant safety AEs, ECG, vital signs, laboratory assessments up to 72 h post dose) and PK data (up to 24 h post-dose for Part A & Part B and 10 days for Part C) will be produced on behalf of the Principal Investigator. Planned doses may be modified following a review of emerging data. Progression to the next SAD dose level and dose selection will be based on the available safety and PK data from at least 6 evaluable participants from the preceding dose level. Progression to the next MAD dose level and dose selection will be based on the available safety and PK data from at least 6 evaluable participants from the preceding dose level. An evaluable participant is defined as a participant who has received the planned dose (active or placebo) and has sufficient PK samples to estimate  $C_{max}$  and  $AUC_{0.24}$ . Dose escalation will be dependent upon generation of acceptable safety (and PK) data. If it is not appropriate to escalate the dose according to the proposed dose escalation schedule, then the same dose, an intermediate dose or a lower dose may be given following discussion between the Sponsor and the Principal Investigator (or deputy) if no stopping criteria are met.

Outputs for the safety review will be presented as Excel listings of the clinical database.

# 8 INTERIM ANALYSES

Other than data review for dose escalation purposes (see section 7), no interim PKor safety analyses are planned for this study.

# 9 DATA

#### 9.1 ECRF DATA

Data captured in the eCRF will be provided by Simbec-Orion Data Management to the Statistics department as SAS datasets in a standard format. Study Data Tabulation Model (SDTM) datasets will be derived from the raw database and Analysis Data Model (ADaM) from SDTM. Both SDTM and ADaM domains will be used for programming the outputs to be included in the Clinical Study Report (CSR). Specifications of both SDTM and ADaM will be provided in a separate document. SDTM/ADaM programming will begin when populated SAS datasets are available.

#### 9.2 EXTERNAL DATA

# 9.2.1 Laboratory Data

Transfers of safety laboratory data will be provided by Simbec-Orion Laboratory Services, delivered to Simbec-Orion Data Management via electronic transfer and stored within the study database and subsequently, within the appropriate SDTM and ADaM domains.. Details of laboratory data are documented in the Data Management Plan (DMP). Populated test transfers will be received before programming can start.





The following results will be included:

- Hematology: Hemoglobin, hematocrit, mean corpuscular volume, mean corpuscular hemoglobin, mean corpuscular hemoglobin concentration, platelet count, red blood cell count, red blood cell distribution width, white blood cell count and WBC differential count (neutrophils, lymphocytes, monocytes, eosinophils, and basophils) (reported in absolute and percentage values).
- **Biochemistry:** Alanine transaminase, albumin, alkaline phosphatase, aspartate transaminase, bicarbonate, total bilirubin, direct bilirubin (if total bilirubin is raised), calcium, chloride, creactive protein, creatine kinase, creatinine, glucose (random), gamma glutamyltransferase, potassium, total protein, sodium, urea, total serum testosterone and luteinizing hormone.
- **Urinalysis:** Bilirubin, blood, glucose, ketones [or ketone bodies], leucocytes, nitrite, pH, protein, specific gravity, and urobilinogen.
- Coagulation: International normalized ratio, Activated partial thromboplastin time and prothrombin time.
- **Microscopy:** In the event that the urinalysis 'dipstick' test result is positive for nitrite and/or 2+ or more reported for protein, blood, and/or leucocytes, the following test parameters will be reported microscopically: bacteria, casts (non-pathogenic), casts (pathogenic), crystals, epithelial cells, red blood cells and white blood cells
- Virology: HBsAg, HCV Ab and HIV test (antibodies to HIV-I and HIV-2).
- COVID-19 Test: A nasopharyngeal and/or oropharyngeal swab will be collected. COVID-19
  testing will be routinely performed via lateral flow test (LFT) however, a RT-PCR test may be
  performed at the Pl's discretion.
- **Drugs of Abuse Screen and Alcohol:** alcohol, amphetamines, barbiturates, benzodiazepines, cannabinoids/tetrahydrocannabinoids (THC), cocaine, cotinine, methadone, and opiates.
- Other Parameters: Any further parameters that are taken at the request of the Investigator that are not included as part of the above categories will be included in an 'Other Laboratory Data' listing.

### 9.2.2 Other non-CRF data

### Pharmacokinetic Data

Plasma and urine AX-158 concentration data will be delivered to Simbec-Orion Data Management via electronic transfer from Simbec-Orion Laboratory Services and stored as a SAS dataset. This data will be stored in the appropriate SDTM domain and subsequent ADaM domain and will be used to produce the file provided to the pharmacokinetic team in order to derive the pharmacokinetic parameters using Phoenix WinNonlin v8.3 or higher. Derived PK parameters will be received from the PK Analyst as a SAS .xpt file in an agreed format and stored in the appropriate SDTM and ADaM domains.



#### 9.3 RANDOMISATION LIST

The randomisation list (in SAS dataset format) will be released following DBL and incorporated into the relevant SDTM/ADaM domains.

#### 9.4 PROGRAMMING AND DATA REVIEW

Programming of datasets, tables, figures and listings will be ongoing while study data management activities are in progress.

Prior to DBL, a review of the clinical database will be conducted. Outputs for the data review will be produced as Excel outputs of the clinical database. A DRM will be held to discuss the outcome of this review, any potential impact on the analyses, analysis sets and protocol deviations. Meeting minutes will be created which will include details of decisions surrounding analysis sets and protocol deviation classification. Once all data issues have been resolved, the analysis sets approved and protocol deviation classifications agreed, the database will be locked. The post-lock SDTM/ADaM datasets will be generated, the TFLs will be run and quality control (QC) will take place.

# 10 STATISTICAL METHODS

#### 10.1 GENERAL PRINCIPLES

- All statistical methods will be based on the International Conference on Harmonisation (ICH) E9 document "Statistical Principles for Clinical Trials".
- All data collected will be presented within data listings.
- Generally, for Part A and Part C, data listings will be sorted by subject, visit and treatment, with the exception of baseline data listings which will be sorted by treatment, subject and visit.
- Generally, for Parts A and C, data listings will be sorted by part, cohort, treatment, subject, visit/time point. Generally, for Part B, data listings will be sorted by part, subject, visit and treatment, where appropriate.
- Generally, data will be summarised by treatment for each part separately. Where appropriate, a summary of all active treatments (Parts A and C) and treatments overall will be included. For Part B, baseline data will be summarised overall. The format of the summaries is defined in the shells at the end of this document.
- Repeated visits will be denoted with 'RPT'. Unscheduled visits will be denoted with 'UNS'.
- In summary and analysis tables of continuous variables, standard descriptive statistics (N [number within analysis set, or group, or subgroup], n [number of observations included in analysis], mean, standard deviation [SD], median, minimum and maximum) will be presented. Least squares means (LSMean) and 90/95% confidence intervals (CI) will be presented in the statistical analysis outputs as appropriate. For PK summaries, geometric mean and coefficient of variation (%CV) will also be used to summarise the data.
- Unless otherwise specified, the minimum and maximum statistics will be presented in summary tables to the same number of decimal places as the original data. The mean, median, LSMean, and CI will be presented to one more decimal place than the original data. SD will be presented to two more decimal places than the original data.
- Derived PK parameters and concentration data listings and summaries will be presented to 3 significant figures (with the exception of CV%, which will be presented to 1 decimal place). The


Document Title: SAP Template - Phase 1

Document Number: TEMP-00109
Previous Document Number: STATt008





ratio of the geometric LSMeans (i.e. test/reference) and its associated confidence interval will be presented to 2 decimal places.

- In summary tables of categorical variables, the number of non-missing observations by category will be presented along with percentages. Unless otherwise specified, the denominator for each percentage will be the number of non-missing observations.
- All percentages will be presented to one decimal place.
- P-values will be rounded to four decimal places. P-values less than 0.0001 will be reported as <0.0001 in tables.</li>
- All plots will use a linear time scale for the nominal times of the visits and will be labelled by time point.
- For post-dose assessments, only data obtained from scheduled visits/time points will be used in summary tables. Post-dose repeat or unscheduled assessments will be listed only. For assessments occurring prior to dosing (i.e. Screening, Day -1, Day 1 pre-dose), the last repeat assessment for each visit will be included in the summary tables and, where repeats of baseline values occur, the last assessment will be used to calculate change from baseline.
- Dates and times for all output presentations will be presented in ISO 8601 Datetime format.
- All outputs will present data in a format that complies with CDISC required terminology and codelists and the SAP will use American-English spelling in line with CDISC terminology, where appropriate (i.e. hematology).
- All statistical analysis will be performed using SAS EG 8.3 or higher.
- All hypothesis testing will be carried out at the 5% (2-sided) significance level unless stated otherwise.
- Generally, character values will be left aligned and numeric values will be decimally aligned.
- If no data is available for a specific output, the output will be produced stating an appropriate message indicating no data was present.
- If any issues arise with the planned analysis of the final data, alternative statistical methods may be used and any changes documented in the statistical methods section of the clinical study report (CSR), including the rationale for use.
- With the exception of PK data, for numeric data which includes non-numeric values (e.g. laboratory results reported as <10 or >100), results reported as  $< x \le x$ ,  $\ge x > x$  will be treated as x for inclusion within the summaries/statistical analysis but will listed as reported. Refer to section 11.4 for handling of non-numeric PK data.

## 10.2 STRATIFICATION AND COVARIATE ADJUSTMENT

None.

### 10.3 INTERACTIONS

None.

#### 10.4 MISSING DATA

No methods to account for missing safety data will be used.

Version:
Document Title:
Document Number:
Previous Document Number:

3.0 SAP Template - Phase 1 TEMP-00109 STATt008





In the instance of missing pharmacokinetic blood samples, the trapezoidal rule will be employed between the samples immediately before and after the missing sample for the AUC calculations.

#### 10.5 POOLING OF SITES

Not applicable.

#### 10.6 MULTIPLE COMPARISONS

No multiplicity adjustments are planned.

### 10.7 SUBGROUP ANALYSES

None.

# 10.8 STATISTICAL ISSUES

None.

# 11 STATISTICAL OUTPUT

General principles for layout of the statistical output are described in Section 10.1. Layout and specifications are illustrated for each unique table in the table shells in Section 14.

#### 11.1 SUBJECT DISPOSITION

The subject disposition table will summarise the following data:

- The number of consented subjects
- The number of subjects receiving each treatment
- The number (%) of subjects who completed/withdrew from the study and the associated reasons for withdrawal
- The number (%) of subjects in each analysis set

All percentages will be calculated from the number of dosed subjects within a treatment group for Parts A and C or number of dosed subjects for Part B.

Screening and study completion/termination data (including informed consent information) will also be listed. A listing of all protocol deviations will be presented including major/minor classification. A data listing presenting subject eligibility for each analysis set and the reason for exclusion from an analysis set will also be presented.

Disposition data will be listed and summarised for the All Consented Set.


**Document Title:**SAP Template - Phase 1 **Document Number:**TEMP-00109

**Previous Document Number:** 

STATt008



#### 11.2 SUBJECT CHARACTERISTICS AT BASELINE

# 11.2.1 Demographic and Baseline Characteristics

Demographic data will be listed. Descriptive statistics (number of participants in the analysis set (N), number of participants with non-missing observations (n), mean, standard deviation (SD), minimum, median, and maximum) will be tabulated for the continuous variables age, height, weight and BMI at Screening and frequencies (number and %) for the categorical variables race and ethnicity.

Demographic data will be listed and summarised using the Safety Set.

### 11.3 EFFICACY ANALYSES

Not applicable.

#### 11.4 PK ANALYSES

#### 11.4.1 Concentration Data

Plasma PK samples will be collected for the measurement of AX-158 at the following time points:

## Part A:

- Day I pre-dose, 30 mins, 45 mins, Ih, 2h, 3h, 4h, 6h, 8h, 12h
- Day 2: 24h, 36h
- Day 3: 48h
- Day 4: 72h

## **Part B:** For both treatment periods

- Day I pre-dose, 30 mins, 45 mins, 1h, 2h, 3h, 4h, 6h, 8h, 12h
- Day 2: 24h, 36h
- Day 3: 48h
- Day 4: 72h

#### Part C:

- Day I and Day I0 pre-dose, Ih, 2h, 3h, 4h, 5h, 6h, 8h, I2h
- Day 2 and Day 11: 24h, 36h
- Day 3 and Day 12: 48h
- Day 4 and Day 13: 72h
- Day 5: pre-dose
- Day 6: Pre-dose
- Day 7: Pre-dose
- Day 8: Pre-dose

Plasma AX-158 concentrations will be listed along with blood sampling times and details of any sampling time deviations and summarised for each treatment using the descriptive statistics N, n, arithmetic mean,

Version:

**Document Title:** SAP Template - Phase 1

TEMP-00109 **Document Number:** STATt008



geometric mean, arithmetic standard deviation (SD), coefficient of variation (CV%), minimum, median and maximum.

The individual subject plasma AX-158 concentration profiles over time will be presented graphically on both linear and semi-logarithmic scales with each subject on a separate plot. For Part C, Day I and Final Dosing Day (Day 10) profiles will be presented on the same plot. The geometric mean plasma AX-158 concentration profiles over time will be presented graphically on both linear and semi-logarithmic scales with all treatments on the same plot, with separate plots for Day I and Final Dosing Day profiles for Part C.

<u>Urine PK</u> samples will be collected for the measurement of AX-158 at the following time intervals: pre-dose and in intervals of 0-12, 12-24, 24-48 and 48-72 h post-dose on Day I and Day I0.

Urine AX-158 concentrations will be listed along with urine volumes and summarised for each treatment using the descriptive statistics N, n, arithmetic mean, geometric mean, arithmetic standard deviation (SD), coefficient of variation (CV%), minimum, median and maximum.

For inclusion within the summary tables and plots, plasma and urine concentrations below the lower limit of quantification (LLOQ) will be imputed as zero at pre-dose and as LLOQ/2 for post-dose samples. They will be listed as recorded. Data reported as not reportable or no sample/result will be handled as missing (i.e. no assumption will be made about the actual concentration).

For inclusion within the summary tables and figures, when calculating the geometric mean concentrations at pre-dose where zero values are likely to be observed, a small value (e.g. 0.001 or smaller) will be added to all individual subject pre-dose concentration values prior to calculation of the mean. This value will then be subtracted after back-transformation, i.e.

$$\textit{Geometric Mean} = \exp(\frac{1}{n} \sum_{n=1}^n \log(x_i + 0.001)) - 0.001$$
 where  $x_i$  are the individual concentration values at pre-dose.

This method is only required for pre-dose results as zero values will not occur for post-dose time points (due to the above imputation method of BLQ values). For post-dose time points, the geometric mean will be calculated using the standard formula:

Geometric Mean = 
$$\exp(\frac{1}{n}\sum_{n=1}^{n}\log(x_i))$$
.

Concentration data listings and individual plots will be presented using the Safety Set. Concentration data summaries and mean plots will be presented using the PK Set. All concentration data included in listings and summaries will be presented to 3 significant figures.

#### 11.4.2 Derived PK Parameters

The derived pharmacokinetic parameters of plasma AX-158 will be determined from the individual concentration versus time data using WinNonlin Phoenix v8.3 or higher. The actual time of blood sample will be used in the calculation of the derived PK parameters. Should the actual time be unavailable but a blood sample was taken, the nominal time point will be assigned.

For the purpose of calculating PK parameters, BLQ values will be imputed as zero at pre-dose and set to missing for post-dose time points. If a Day I, pre-dose result is missing, it will be imputed as zero. The following plasma AX-158 PK parameters will be calculated using standard non-compartmental methods:

Version: **Document Title: Document Number:** 

**Previous Document Number:** 

SAP Template - Phase 1 TEMP-00109 STATt008



# Part A:

| Pharmacokinetic<br>Parameter and<br>Unit | Definition | Computation | WinNonlin<br>Parameter<br>Name |
|---|---|---|---|
| C <sub>max</sub> (µg/mL) | Maximum concentration. | Maximum observed concentration, occurring at Tmax. If not unique, then the first maximum is used. | Cmax |
| T <sub>max</sub> (h) | The time to maximum observed concentration. | Time of maximum observed concentration. If the maximum observed concentration is not unique, then the first maximum is used. | Tmax |
| λ <b>z (I/h)</b> | Elimination rate constant. | First order rate constant associated with the terminal (log-linear) portion of the curve. Estimated by linear regression of time vs. log concentration; the regression analysis should contain data from at least 3 different time points in the terminal phase | lambda_z |
| t <sub>1/2</sub> (h) | Terminal elimination half-life. | $=\ln(2)/\lambda z$ | HL_Lambda_z |
| AUC <sub>0-24</sub> (h*μg/mL) | Area under the concentration-time curve (AUC) from the time of dosing to 24 h post-dose | AUC measured from the concentration at time of dosing to 24 hours post dose. The AUC is computed using the linear up-log down trapezoidal rule. | AUC0-24 |
| AUC <sub>0-t</sub> (h*µg/mL) | Area under the concentration-time curve (AUC) from the time of dosing to the time of the last measurable concentration. | AUC measured from the concentration at time of dosing to the last measurable positive concentration. The AUC is computed using the linear up-log down trapezoidal rule. | AUClast |
| AUC <sub>0-inf</sub> (h*µg/mL) | AUC extrapolated to infinity. | AUC measured from the concentration at time of dosing extrapolated to infinity based on the last observed concentration. | AUCINF_obs |

Version: Document Title: Document Number: Previous Document Number:

SAP Template - Phase 1 TEMP-00109 STATt008



| Pharmacokinetic<br>Parameter and<br>Unit | Definition | Computation | WinNonlin<br>Parameter<br>Name |
|---|---|---|---|
| | | $= AUC_{0-t} + \frac{C_{lastobs}}{\lambda z}$ | |
| AUC <sub>%extrap.</sub> (%) | Percentage of AUC <sub>0-inf</sub> due to extrapolation from last observed concentration to infinity. | Percentage of AUC <sub>0-inf</sub> due to extrapolation from time of last measurable positive concentration to infinity. $= \frac{AUC_{0-inf} - AUC_{0-t}}{AUC_{0-inf}} \cdot 100$ | AUC_%Extrap<br>_obs |
| CL/F (L/h) | Apparent total body clearance, calculated as Dose / AUC <sub>0-inf</sub> . | $= Dose/AUC_{0-inf}$ | CL_F_obs |
| Vz/F (L) | Apparent Volume of Distribution during the terminal phase. | $= \frac{Dose}{\lambda z. AUC_{0-inf}}$ | Vz_F_obs |
| \(\lambda z \text{ lower}\) (listed only) | Elimination rate constant lower limit. | Lower limit on Time for values to be included in the calculation of $\lambda z$ | Lambda_z_lower |
| Az upper<br>(listed only) | Elimination rate constant upper limit. | Upper limit on Time for values to be included in the calculation of $\lambda z$ | Lambda_z_upper |
| No. points λz (listed only) | Number of points used for elimination rate constant. | Number of points used for elimination rate constant | No_points_<br>Lambda_z |
| R <sup>2</sup> adjusted<br>(listed only) | R <sup>2</sup> adjusted. | Goodness of fit statistic for the terminal elimination phase, adjusted for the number of points used in the estimation of $\lambda z$ | Rsq_adjusted |

# Part B

| Pharmacokinetic<br>Parameter and<br>Unit | Definition | Computation | WinNonlin<br>Parameter<br>Name |
|---|---|---|---|
| C <sub>max</sub> (µg/mL) | Maximum concentration. | Maximum observed concentration, occurring at | Cmax |


Document Title: SAP Template - Phase 1
Document Number: TEMP-00109
Previous Document Number: STATt008





| Pharmacokinetic<br>Parameter and<br>Unit | Definition | Computation | WinNonlin<br>Parameter<br>Name |
|---|---|---|---|
| | | Tmax. If not unique, then the first maximum is used. | |
| T <sub>max</sub> (h) | The time to maximum observed concentration. | Time of maximum observed concentration. If the maximum observed concentration is not unique, then the first maximum is used. | Tmax |
| T <sub>lag</sub> (h) | The delay in achieving<br>Tmax | Time of observation prior to the first observation with a measurable (non-zero) concentration. | Tlag |
| λ <b>z</b> (1/h) | Elimination rate constant. | First order rate constant associated with the terminal (log-linear) portion of the curve. Estimated by linear regression of time vs. log concentration; the regression analysis should contain data from at least 3 different time points in the terminal phase | lambda_z |
| t <sub>1/2</sub> (h) | Terminal elimination half-life. | $=\ln(2)/\lambda z$ | HL_Lambda_z |
| AUC <sub>0-24</sub> (h*μg/mL) | Area under the concentration-time curve (AUC) from the time of dosing to 24 h post-dose | AUC measured from the concentration at time of dosing to 24 hours post dose. The AUC is computed using the linear up-log down trapezoidal rule. | AUC0-24 |
| AUC <sub>0-t</sub> (h*μg/mL) | Area under the concentration-time curve (AUC) from the time of dosing to the time of the last measurable concentration. | AUC measured from the concentration at time of dosing to the last measurable positive concentration. The AUC is computed using the linear up-log down trapezoidal rule. | AUClast |
| AUC <sub>0-inf</sub> (h*µg/mL) | AUC extrapolated to infinity. | AUC measured from the concentration at time of dosing extrapolated to infinity based on the last observed concentration. | AUCINF_obs |

Version:
Document Title:
Document Number:
Previous Document Number:

SAP Template - Phase 1 TEMP-00109 STATt008



| Pharmacokinetic<br>Parameter and<br>Unit | Definition | Computation | WinNonlin<br>Parameter<br>Name |
|---|---|---|---|
| | | $= AUC_{0-t} + \frac{C_{lastobs}}{\lambda z}$ | |
| AUC <sub>%extrap.</sub> (%) | Percentage of AUC <sub>0-inf</sub> due to extrapolation from last observed concentration to infinity. | Percentage of AUC <sub>0-inf</sub> due to extrapolation from time of last measurable positive concentration to infinity. $= \frac{AUC_{0-inf} - AUC_{0-t}}{AUC_{0-inf}} \cdot 100$ | AUC_%Extrap<br>_obs |
| CL/F (L/h) | Apparent total body clearance, calculated as Dose / AUC <sub>0-inf</sub> . | $= Dose/AUC_{0-inf}$ | CL_F_obs |
| Vz/F (L) | Apparent Volume of Distribution during the terminal phase. | $= \frac{Dose}{\lambda z. AUC_{0-inf}}$ | Vz_F_obs |
| λz lower<br>(listed only) | Elimination rate constant lower limit. | Lower limit on Time for values to be included in the calculation of $\lambda z$ | Lambda_z_lower |
| λz <sub>l</sub> upper<br>(listed only) | Elimination rate constant upper limit. | Upper limit on Time for values to be included in the calculation of $\lambda z$ | Lambda_z_upper |
| No. points λz (listed only) | Number of points used for elimination rate constant. | Number of points used for elimination rate constant | No_points_<br>Lambda_z |
| R <sup>2</sup> adjusted<br>(listed only) | R <sup>2</sup> adjusted. | Goodness of fit statistic for the terminal elimination phase, adjusted for the number of points used in the estimation of $\lambda z$ | Rsq_adjusted |

# Part C on Day I:



| Pharmacokinetic<br>Parameter and<br>Unit | Definition | Computation | WinNonlin<br>Parameter<br>Name |
|---|---|---|---|
| C <sub>max</sub> (µg/mL) | Maximum concentration. | Maximum observed concentration, occurring at Tmax. If not unique, then the first maximum is used. | Cmax |
| T <sub>max</sub> (h) | The time to maximum observed concentration. | Time of maximum observed concentration. If the maximum observed concentration is not unique, then the first maximum is used. | Tmax |
| AUC <sub>0-24</sub> (h*μg/mL) | Area under the concentration-time curve (AUC) from the time of dosing to 24 h post-dose | AUC measured from the concentration at time of dosing to 24 hours post dose. The AUC is computed using the linear up-log down trapezoidal rule. | AUC0-24 |
| AUC <sub>0-tau</sub> (h*µg/mL) (only required if non-q.d. dosing regimen) | Area under the plasma concentration-time curve (AUC) from the time of dosing to <x> hours (dosing interval) after the Day <x> dose.</x></x> | AUC measured from the concentration at time of dosing to the concentration at <x> hours. The AUC is computed using the linear up-log down trapezoidal rule.</x> | AUC_TAU |

# Part C on Final Dosing Day:

| Pharmacokinetic<br>Parameter and<br>Unit | Definition | Computation | WinNonlin<br>Parameter<br>Name |
|---|---|---|---|
| C <sub>max</sub> (µg/mL) | Maximum concentration. | Maximum observed concentration, occurring at Tmax. If not unique, then the first maximum is used. | Cmax |
| T <sub>max</sub> (h) | The time to maximum observed concentration. | Time of maximum observed concentration. If the maximum observed concentration is not unique, then the first maximum is used. | Tmax |



| Pharmacokinetic<br>Parameter and<br>Unit | Definition | Computation | WinNonlin<br>Parameter<br>Name |
|---|---|---|---|
| λ <b>z</b> (I/h) | Elimination rate constant. | First order rate constant associated with the terminal (log-linear) portion of the curve. Estimated by linear regression of time vs. log concentration; the regression analysis should contain data from at least 3 different time points in the terminal phase | lambda_z |
| t <sub>1/2</sub> (h) | Terminal elimination half-life. | $= \ln(2)/ \lambda z$ | HL_Lambda_z |
| AUC <sub>0-24</sub> (h*µg/mL) | Area under the concentration-time curve (AUC) from the time of dosing to 24 h post-dose | AUC measured from the concentration at time of dosing to 24 hours post dose. The AUC is computed using the linear up-log down trapezoidal rule. | AUC0-24 |
| AUC <sub>0-tau</sub> (h*µg/mL) (only required if non-q.d. dosing regimen) | Area under the plasma concentration-time curve (AUC) from the time of dosing to 24 hours (dosing interval) after the Day 10 dose. | AUC measured from the concentration at time of dosing to the concentration at 24 hours. The AUC is computed using the linear up-log down trapezoidal rule. | AUC_TAU |
| AUC <sub>0-t</sub> (h*μg/mL) | Area under the concentration-time curve (AUC) from the time of dosing to the time of the last measurable concentration. | AUC measured from the concentration at time of dosing to the last measurable positive concentration. The AUC is computed using the linear up-log down trapezoidal rule. | AUClast |
| AUC <sub>0-inf</sub> (h*µg/mL) | AUC extrapolated to infinity. | AUC measured from the concentration at time of dosing extrapolated to infinity based on the last observed concentration. $= AUC_{0-t} + \frac{C_{lastobs}}{\lambda z}$ | AUCINF_obs |
| AUC <sub>%extrap.</sub> (%) | Percentage of AUC <sub>0-inf</sub> due to extrapolation from last observed | Percentage of AUC <sub>0-inf</sub> due to extrapolation from time of last measurable positive concentration to infinity. | AUC_%Extrap<br>_obs |

Version:3Document Title:SDocument Number:TPrevious Document Number:S

SAP Template - Phase 1 TEMP-00109 STATt008



| Pharmacokinetic<br>Parameter and<br>Unit | Definition | Computation | WinNonlin<br>Parameter<br>Name |
|---|---|---|---|
| | concentration to infinity. | $= \frac{AUC_{0-inf} - AUC_{0-t}}{AUC_{0-inf}} \cdot 100$ | |
| CL/F (L/h) | Apparent total body clearance, calculated as Dose / AUC <sub>0-inf</sub> . | $= Dose/AUC_{0-inf}$ | CL_F_obs |
| Vz/F (L) | Apparent Volume of Distribution during the terminal phase. | $= \frac{Dose}{\lambda z. AUC_{0-inf}}$ | Vz_F_obs |
| \(\lambda z \text{ lower}\) (listed only) | Elimination rate constant lower limit. | Lower limit on Time for values to be included in the calculation of $\lambda z$ | Lambda_z_lower |
| λz upper<br>(listed only) | Elimination rate constant upper limit. | Upper limit on Time for values to be included in the calculation of $\lambda z$ | Lambda_z_upper |
| No. points λz (listed only) | Number of points used for elimination rate constant. | Number of points used for elimination rate constant | No_points_<br>Lambda_z |
| R <sup>2</sup> adjusted<br>(listed only) | R <sup>2</sup> adjusted. | Goodness of fit statistic for the terminal elimination phase, adjusted for the number of points used in the estimation of $\lambda z$ | Rsq_adjusted |

The terminal elimination rate constant ( $\lambda z$ ) will be calculated by log-linear regression of the terminal portion of the concentration-time curve only where there are sufficient data i.e. at least 3 time points excluding  $C_{max}$  and adjusted  $R^2$  is greater than or equal to 0.85; lower adjusted  $R^2$  values may be acceptable at the discretion of the PK analyst if the elimination phase is clearly defined by the profile, values lower than 0.85 will be flagged within the data listing. If these criteria are not fulfilled, parameters dependent on  $k_{el}$  for calculation will not be reported.

The following urine PK parameters will be calculated:

# Part C on Day I and Final Dosing Day

Version:
Document Title:
Document Number:
Previous Document Number:

SAP Template - Phase 1 TEMP-00109 STATt008



| Pharmacokinetic<br>Parameter and<br>Unit | Definition | Computation | WinNonlin<br>Parameter Name |
|---|---|---|---|
| Ae (µg) | Cumulative amount of study drug excreted in urine during a time interval. | The sum of the individual urine volume * urine concentration of study drug. $= \Sigma \ (Concentration \ . Volume)$ | N/A (calculated using SAS) |
| Ae% (%) | Percentage of study drug excreted in urine during a time interval. | = 100 . Ae/Dose | N/A (calculated using SAS) |
| CL <sub>R</sub> (L/h) | Renal clearance. | $= Ae/AUC_{0-t}$ | N/A (calculated using SAS) |

The derived urine pharmacokinetic parameters Ae, Ae%, CumAe, CumAe%, CLR will be determined from the individual urine concentration versus time data using SAS EG v8.3 or higher.

Derived PK parameters will be listed along with the points used to calculate  $\lambda z$  (lower, upper, and number used) and coefficient of determination (R²) adjusted. The derived PK parameters will also be summarised. The descriptive statistics presented will be N, n, arithmetic mean, geometric mean (with the exception of  $T_{max}$ ), SD, coefficient of variation (CV%), minimum, median, and maximum. Any AUC<sub>% extrap</sub> values greater than 20% will be flagged within the data listing. In accordance with regulatory guidance, the associated data should not be excluded from analysis but if this is observed for

>20% of the profiles, the validity of the study may be in question.

In the instance of a significant sample time deviation ( $\geq$  5% of nominal time i.e. 72 min) for the 24 h PK sample, the AUC<sub>0-24</sub> values will be excluded from statistical analysis, but will be calculated, included in the derived PK data listing and flagged. Where a non-significant sample time deviation ( $\leq$ 72 min) for the 24 h PK sample occurs and the terminal elimination rate constant (lambda\_z) is estimable, this will be used to estimate AUC<sub>0-24</sub>. Where a non-significant sample time deviation ( $\leq$  72 min) for the 24 h PK sample occurs and the terminal elimination rate constant (lambda\_z) is not estimable, WNL is unable to estimate AUC<sub>0-24</sub>. Therefore, in order for an AUC<sub>0-24</sub> value to be estimated, the actual sampling time (including bleed time deviations) at the 24 h nominal time point will be used for the partial AUC settings.

PK parameter listings will be presented using the Safety Set. PK parameter summaries will be presented using the PK Set. All PK parameter data included in listings and summaries will be presented to 3 significant figures (with the exception of CV% which will be presented to one decimal place).

### 11.4.3 Statistical Analysis of PK Data

# **Dose Proportionality**

Dose proportionality will be assessed by performing a regression analysis of the log-transformed  $C_{max}$ ,  $AUC_{0-t}$ ,  $AUC_{0-24}$  and  $AUC_{0-inf}$  values versus the log-transformed dose using the power model with a fixed


Document Title:SAP Template - Phase 1Document Number:TEMP-00109Previous Document Number:STATt008



effect for log(dose). For each parameter, point estimates for the intercept and the slope of the regression line and the 95% CI of the slope will be calculated. In addition, estimated geometric LSMeans and corresponding 95% CIs will be presented for each dose level.

The power model is defined as:

$$log_e(C_{max}, AUC_{0-t}, AUC_{0-inf}) = \alpha + \beta log_e(Dose) + \varepsilon$$
,

where  $\alpha$  is the intercept,  $\beta$  is the slope and  $\epsilon$  is the error term.

Geometric LSMeans and associated 95% CIs along with individual subject values for the derived pharmacokinetic parameters  $C_{max}$ ,  $AUC_{0-t}$  and  $AUC_{0-inf}$  will be presented graphically versus dose with each parameter presented on a separate plot.

# **Dose Independence**

Dose independence will be assessed for  $t\frac{1}{2}$  and CL/F by performing a regression analysis of the untransformed parameters versus dose with a fixed effect for dose. For each parameter, point estimates for the intercept and the slope of the regression line and the 95% CI of the slope will be calculated. In addition, estimated LSMeans and corresponding 95% CIs will be presented for each dose level.

LSmeans and associated 95% CIs along with individual subject values for the derived pharmacokinetic parameters  $t\frac{1}{2}$  and CL/F will be presented graphically versus dose.

#### 11.4.3.1 Part B - Food Effect

Following logarithmic transformation,  $C_{max}$ ,  $AUC_{0-t}$  and  $AUC_{0-inf}$  values will be subjected to an analysis of variance (ANOVA) including fixed effects for sequence, period, treatment and subject nested within sequence. Point estimates and 90% confidence intervals will be constructed for the contrasts between treatments using the residual mean square error obtained from the ANOVA. The point and interval estimates will be back-transformed to give estimates of the ratios of the geometric LSMeans and corresponding 90% Cls. In addition, estimated geometric LSMeans and corresponding 95% Cls for each treatment and the within-subject CV% will be presented.

The geometric LSMean ratios and corresponding 90% CIs for  $C_{max}$  AUC<sub>0-t</sub> and AUC<sub>0-inf</sub> will be represented graphically (a plot with error bars) with all parameters on one graph. On the same graph, points indicating individual within-subject ratios for the three PK parameters will be presented. Reference lines will be included to indicate the 80.00% and 125.00% CI thresholds.

Each treatment comparison will be analysed separately and will only include data from subjects who are included in the PK Set for the two treatments being evaluated.

#### 11.4.3.2 Part C (MAD) - Dose-Proportionality/Independence

# **Dose-Proportionality**

For Day I and Final Dosing Day (Day 10), dose proportionality will be assessed by performing a regression analysis of the log-transformed  $C_{max}$ ,  $AUC_{0-tau}$  and  $AUC_{0-inf}$  (Day 10 only) values versus the log-transformed dose using the power model with a fixed effect for log (dose). For each parameter, a point estimate and 95 % CI will be calculated for the slope of the regression line.


**Document Title:**SAP Template - Phase 1 **Document Number:**TEMP-00109

Previous Document Number:

STATt008



The power model is defined as:

$$log_e(C_{max}, AUC_{0-t}, AUC_{0-inf}) = \alpha + \beta log_e(Dose) + \epsilon$$

where  $\alpha$  is the intercept,  $\beta$  is the slope and  $\epsilon$  is the error term.

Geometric LSMeans and associated 95% CIs along with individual subject values for the derived pharmacokinetic parameters  $C_{max}$ ,  $AUC_{0-t}$  and  $AUC_{0-inf}$  will be presented graphically versus dose with each parameter presented on a separate plot.

# **Dose Independence**

For Final Dosing Day (Day 10), dose independence will be assessed for  $t\frac{1}{2}$  and CL/F by performing a regression analysis of the untransformed parameters versus dose with a fixed effect for dose. For each parameter, a point estimate and corresponding 95 % CI will be calculated for the slope of the regression line.

#### 11.4.3.3 Part C (MAD) - Steady State

For each treatment, log-transformed trough concentration levels at pre-dose on Day 5 and Final Dosing Day (Day 10) will be subjected to a mixed effects analysis of variance (ANOVA) with study day as a fixed effect and subject as a random effect in order to establish whether steady-state has been attained for each treatment. The point and interval estimates will be back-transformed to give estimates of the ratios of the geometric LSMeans and corresponding 90% Cls for the comparisons of each consecutive day (i.e. Day 10/Day 5). In addition, estimated geometric LSMeans and corresponding 95% Cls will be presented for each study day.

The geometric LSMean ratio and corresponding 90% CI for the Day 10/Day 5 comparison will be presented graphically (a plot with error bars) with all treatments on one graph. On the same graph, points indicating individual within-subject ratios for the comparison will be presented.

## 11.4.3.4 Part C (MAD) - Accumulation

For each dose level, log-transformed  $C_{max}$  and  $AUC_{0-tau}$  (only applicable if non-q.d. dosing regimen is implemented) values on Day I and Final Dosing Day (Day I0) will be subjected to an ANOVA with study day as a fixed effect and subject as a random effect. For comparison, point estimates and 90% Cls for the difference between Day I0 and Day I will be constructed using the residual mean square error obtained from the ANOVA for each dose level. The point and interval estimates will then be back transformed to give estimates of the ratios of the geometric LSMeans and corresponding 90% Cls. In addition, estimated geometric LSMeans and corresponding 95% Cls will be presented for each study day.

The geometric LSMean ratios and corresponding 90% CIs for  $C_{max}$  and  $AUC_{0-tau}$  will be represented graphically (a plot with error bars) with all dose levels on one graph, one graph per parameter. On the same graph, points indicating individual within-subject ratios will be presented.

Statistical analysis of PK parameters will be performed using the PK set.





## 11.5 PD ANALYSES

Not applicable.

#### 11.6 SAFETY ANALYSES

### 11.6.1 Adverse Events

All adverse events (AEs) will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) dictionary version 24.1.

All AEs, including those which occurred prior to the first treatment administration, will be listed. Only treatment emergent adverse events (TEAEs), i.e., existing conditions that worsen or events that occur during the course of the study after administration of study drug, will be included within the summary tables. AEs that occur intermittently will be reported as separate events.

### Part A and Part C:

An AE will be assigned to treatment if it starts on or after dosing. Where there are only partial dates/times recorded for an adverse event, the adverse event will be assigned to treatment if it cannot be ruled out based on the partial information.

#### Part B:

An AE will be assigned to the most recent treatment if it starts on or after the corresponding dose. Where there are only partial dates/times recorded for an adverse event, the adverse event will be assigned to every treatment where it cannot be ruled out based on the partial information.

An overall summary of AEs will be produced including the number of TEAEs; the number and % of subjects reporting at least I TEAE, serious TEAE (where SAE is reported as 'Yes'), TEAE leading to withdrawal from the study (Action recorded as 'Study Drug Discontinued'), TEAE leading to death (Outcome recorded as 'Fatal'); the number and % of subjects reporting TEAEs by severity and relationship to study drug. A subject with multiple occurrences of any AE is counted only once at the maximum level of severity or the strongest relationship to study drug.

The number of TEAEs and the number and % of subjects reporting at least I TEAE will be tabulated by system organ class (SOC) and preferred term (PT). A subject reporting multiple episodes of a particular AE within a treatment period will only contribute I count towards the corresponding SOC and PT.

In order to highlight the most frequently reported TEAEs, the number of TEAEs and the number and % of subjects reporting at least I TEAE will be tabulated by PT in order of descending frequency such that AEs reported by the greatest number of subjects are presented first. A subject reporting multiple episodes of a particular AE will only contribute I count towards the corresponding PT.

In addition, the number and % of subjects reporting TEAEs will be tabulated by maximum severity and strongest relationship to study drug. For the summary of TEAEs by severity, if a subject has multiple events occurring within the same SOC or PT the event with the highest severity will be counted. Similarly, for TEAEs by relationship to study drug, if a subject has multiple events occurring within the same SOC or PT, the event with the strongest relationship to study drug will be counted.

AEs will be listed by treatment. For any adverse event occurring prior to first administration of study drug, treatment will be described as 'Prior to Treatment'.





The derived variables, 'Time from Dose' and 'Duration' will be presented where full date and time are present. If partial dates are present for any parameter required in the calculation, the variable will not be populated. The following will be used to calculate the variables:

**Duration (dd:hh:mm)**: (Date/Time of Resolution - Date/Time of Onset) + I minute;

Time from Dose (dd:hh:mm): (Date/Time of Onset - Date/Time of Start of Dose).

The following will be presented in listing format within the data summaries:

- Serious Adverse Events If there are none present, the listing will be produced stating: 'No subjects experienced any serious adverse events.'.
- Adverse Events which Led to Withdrawal If there are none present, the listing will be produced stating: 'No subjects experienced any adverse events that led to withdrawal.'.
- Adverse Events Leading to Death If there are none present, the listing will be produced stating:
   'No subjects experienced any adverse events that led to death.'.

Adverse event data will be listed and summarised using the Safety Set.

# 11.6.2 Laboratory Data

Routine safety clinical laboratory tests (biochemistry, hematology, coagulation, urinalysis) will be carried out at:

**Part A:** Screening, Day -1, 24h post dose, 72h post dose and at follow-up. An additional urinalysis test will be carried out at Day 1, 12h.

**Part B:** Screening, Day -1, 24h post dose, 72h post dose and at follow-up. An additional biochemistry test will be carried out at Day I pre dose (total serum testosterone only) and an additional urinalysis test will be carried out at Day I - I2h.

<u>Part C:</u> Screening, Day -1, 24h post dose, 72h post dose, pre-dose on Day 5 and at follow-up. An additional biochemistry test (total serum testosterone and LH only) will be carried out at Day 1 pre-dose, Day 5, Day 8 and Day 11 and an additional urinalysis test will be carried out at Day 1, 12h.

The laboratory parameters required for this study are listed in section 9.2.1.

Laboratory data listings will be presented in two ways:

- Out of range values any values that fall outside of the normal/alert ranges based on the reference ranges provided by the Simbec-Orion Laboratory Services (presented in listing format within the data summaries)
- All safety laboratory data (including physician's review (Normal, Abnormal-NCS, Abnormal-CS)) with any out of range values flagged (presented within the data listings).

Descriptive statistics (N, n, mean, SD, minimum, median and maximum) of absolute and change from baseline (last assessment prior to first dose within a treatment period) values for each parameter at each protocol defined time point will be tabulated by treatment.





Microscopy, virology, COVID-19 test, urine drugs of abuse and alcohol screen and any unplanned laboratory parameters will also be listed.

If there are no further parameters databased other than those specified in section 9.2.1 then the 'Other Laboratory Data' listings should display, 'No other laboratory parameters to report'.

Laboratory data will be listed and summarised using the Safety Set.

# 11.6.3 Vital Signs

Vital Signs will be recorded at:

**Part A:** Screening, Day -1, Day 1 pre-dose, 30 mins, 45 mins, 1h, 2h, 3h, 4h, 6h, 8h, 12h, 24h post dose, 36h post dose, 48h post dose, 72h post dose and follow-up.

**Part B:** Screening, Day -1, Day 1 pre-dose, 30 mins, 45 mins, 1h, 2h, 3h, 4h, 6h, 8h, 12h, 24h post dose, 36h post dose, 48h post dose, 72h post dose and follow-up.

<u>Part C:</u> Screening, Day -1, Day 1 and Day 10 at pre-dose, 30 mins, 45 mins, 1h, 2h, 3h, 4h, 6h, 8h, 12h, 24h post dose, 36h post dose, 48h post dose, 72h post dose, pre-dose on Day 5 and follow-up.

A window of ± 10 min in relation to the nominal time-point is allowed.

Vital signs parameters (supine systolic and diasolic blood pressure and pulse rate, oral temperature and respiratory rate) will be listed with any out of normal range values (see Appendix 16.1) flagged (flag appended to relevant result). Descriptive statistics (N, n, mean, SD, minimum, median and maximum) of absolute and change from baseline (Day I, pre-dose [of each treatment period for Part B] or last assessment prior to first dose, as applicable) values at each time point will be tabulated by treatment.

Vitals signs data will be listed and summarised using the Safety Set.

### 11.6.4 Electrocardiogram

12-lead ECGs will be performed at:

Part A: Screening, Day -1, Day 1 pre-dose, 30 min, 4h, 12h, 24h post dose, 48h post dose, 72h post dose, follow-up.

Part B: Screening, Day -1, Day 1 pre-dose, 30 min, 4h, 12h, 24h post dose, 48h post dose, 72h post dose, follow up.

**Part C:** Screening, Day -1, Day 1 and Day 10 at pre-dose, 30 min, 4h, 12h, 24h, 48h, and 72h post dose, pre-dose on Day 5 and follow-up.

A window of  $\pm$  10 min in relation to the nominal time-point is allowed.

12-lead ECG parameters (heart rate, PR interval, QRS width, QT interval and QT interval corrected using Fridericia's formula (QTcF)) will be listed with any out of normal range values (see Appendix 16.1) flagged (flag appended to relevant result). Descriptive statistics (N, n, mean, SD, minimum, median and


**Document Title:**SAP Template - Phase 1 **Document Number:**TEMP-00109

Previous Document Number: Si

STATt008




maximum) of absolute and change from baseline (Day I, pre-dose [of each treatment period for Part B] or last assessment prior to first dose, as applicable) values at each time point will be summarised by treatment.

In addition, frequencies for QTcF data will be calculated and summarised according to the following categories:

#### For absolute values:

- QTc ≤ 450 msec
- 450 < QTc ≤ 480 msec</li>
- 480 < QTc ≤ 500 msec
- QTc > 500 msec.

#### For change from baseline:

- Decreased/No Change
- QTc increase ≤ 30 msec
- 30 < QTc increase ≤ 60 msec
- QTc increase > 60 msec

ECG data will be listed and summarised using the Safety Set.

#### 11.7 OTHER

#### 11.7.1 Prior and Concomitant Medication

Dictionary (WHODD) coding dictionary version September 2021 and listed using the ATC Level 4 class, Preferred Term and verbatim text.

#### Part A and Part C:

A medication will be assigned to treatment if it starts on or after dosing. Where there are only partial dates/times recorded for a medication, the medication will be assigned to treatment if it cannot be ruled out based on the partial information.

#### Part B:

A medication will be assigned to the most recent treatment if it starts on or after the corresponding dose. Where there are only partial dates/times recorded for a medication, the medication will be assigned to every treatment where it cannot be ruled out based on the partial information.

A medication will be regarded as *prior* if it stops prior to first administration of IMP. The treatment phase will be presented as 'Prior to Treatment'. A medication will be regarded as *concomitant* if it starts after dosing or starts before dosing and continues after dosing. For any medication that started prior to first administration of IMP but is ongoing following administration of IMP, the treatment phase will be described as 'Prior and Ongoing'. Otherwise, treatment phase will be described as the treatment the medication started on.

Prior and concomitant medications will be listed by treatment phase using the Safety Set.





#### 11.7.2 All Other Data

All data will be listed using the Safety Set, including the following: Substance Use History, Visit Dates, Medical History, Physical Examination, Inclusion/Exclusion Failures, PD Sampling, IMP Administration and Additional Notes.

#### **Derivations within listings:**

<u>PK blood sampling time deviations</u>: Calculate sample time deviation using actual time – theoretical time, display as minutes.

<u>Analysis sets</u>: Detail whether subject should be included within each of the analysis sets and provide reason for exclusion, as appropriate.

<u>Inclusion/Exclusion criteria</u>: Only failures to be presented. If there are no failures display 'All subjects passed all inclusion/exclusion criteria.'

<u>Protocol deviations</u>: Major/minor classification to be assigned and confirmed by Sponsor.

### 12 VALIDATION

All tables, figures and listings will be subject to independent quality control and visual review and will be independently programmed. Findings will be documented in an Output Summary file quality control form and actions taken will also be documented.

The study summary sheet of the Output Summary file will be completed and signed by all persons who performed programming and QC. The final signed version of the Output Summary will be stored in the electronic Trial Master File (eTMF).

## 13 LITERATURE CITATIONS/REFERENCES

None.



## 14 LIST OF TABLES, FIGURES AND LISTINGS

## List of Tables and Figures Contained in Report Section 14

## 14.1 Disposition and Demographic Data

### 14.1.1 Disposition Data

| Table 14.1.1.1 | Summary of Study Disposition | All Consented<br>Set |
|---|---|---|
| 14.1.2 Demogra | aphic Data and Baseline Characteristics | |
| Table 14.1.2.1 | Summary of Demographic Information | Safety Set |

## 14.2 Efficacy Data

Not applicable.

### 14.3 Safety Data

### 14.3.1 Adverse Events

| Table 14.3.1.1 | Summary of Treatment Emergent Adverse Events | Safety Set |
|---|---|---|
| Table 14.3.1.2 | Summary of Treatment Emergent Adverse Events by System<br>Organ Class and Preferred Term | Safety Set |
| Table 14.3.1.3 | Summary of Treatment Emergent Adverse Events by Preferred Term | Safety Set |
| Table 14.3.1.4 | Summary of Treatment Emergent Adverse Events by System Organ Class, Preferred Term and Severity | Safety Set |
| Table 14.3.1.5 | Summary of Treatment Emergent Adverse Events by System Organ Class, Preferred Term and Relationship to Study Drug | Safety Set |
| Table 14.3.1.6 | Serious Adverse Events | Safety Set |
| Table 14.3.1.7 | Adverse Events Leading to Withdrawal | Safety Set |
| Table 14.3.1.8 | Adverse Events Leading to Death | Safety Set |

#### 14.3.2 Laboratory Safety

| T 1.5.2 Laborato | a y Sarety | |
|---|---|---|
| Table 14.3.2.1 | Biochemistry Out of Normal Range Data | Safety Set |
| Table 14.3.2.2 | Hematology Out of Normal Range Data | Safety Set |
| Table 14.3.2.3 | Coagulation Out of Normal Range Data | Safety Set |
| Table 14.3.2.4 | Urinalysis Out of Normal Range Data | Safety Set |
| Table 14.3.2.5 | Summary of Absolute and Change from Baseline Biochemistry Results | Safety Set |
| Table 14.3.2.6 | Summary of Absolute and Change from Baseline Hematology Results | Safety Set |


 Document Title:
 SAP Template - Phase 1

 Document Number:
 TEMP-00109

 Previous Document Number:
 STATt008





| Table 14.3.2.7 Summary of Absolute and Change from Baseline Coagulation Safety Set Data |
|---|
|---|

### 14.3.3 Vital Signs

| Table 14.3.3.1 | Summary of Absolute and Change from Baseline Vital Signs<br>Data | Safety Set |
|---|---|---|
| 14.3.4 ECG ( | | |
| Table 14.3.4.1 | Summary of Absolute and Change from Baseline 12-lead ECG Data | Safety Set |
| Table 14.3.4.2 | Summary of 12-lead ECG QTcF Categories | Safety Set |

#### 14.4 Pharmacokinetics

#### 14.4.1 Concentration Data

| Table 14.4.1.1 | Summary of Plasma AX-158 Concentration Data | PK Set |
|---|---|---|
| Figure 14.4.1.1 | Geometric Mean Plasma AX-I58 Concentration-Time Curves on a Linear Scale | PK Set |
| Figure 14.4.1.2 | Geometric Mean Plasma AX-158 Concentration-Time Curves on a Semi-Logarithmic Scale | PK Set |

#### 14.4.2 Derived Pharmacokinetics

| Table 14.4.2.1 | Summary of Derived Plasma AX-158 Pharmacokinetic Parameters | PK Set |
|---|---|---|
| Table 14.4.2.2 | Summary of Statistical Analysis of Plasma AX-158 Pharmacokinetic Data - Dose Proportionality | PK Set |
| Table 14.4.2.3 | Summary of Statistical Analysis of Plasma AX-158 Pharmacokinetic Data - Dose Independence | PK Set |
| Figure 14.4.2.1 | Dose Response of Plasma AX-158 Derived Pharmacokinetic Data | PK Set |
| Table 14.4.2.4 | Summary of Statistical Analysis of Plasma AX-158 Pharmacokinetic Data - Food Effect | PK Set |
| Figure 14.4.2.2 | Food Effect Least Squares Geometric Mean Ratios and 90% Cls of Plasma AX-158 PK Data | PK Set |
| Table 14.4.2.5 | Summary of Statistical Analysis of Plasma AX-158 Pharmacokinetic Data - Steady State | PK Set |
| Figure 14.4.2.3 | Steady State Least Squares Geometric Mean Ratios and 90% Cls of Plasma AX-158 Concentration Data | PK Set |
| Table 14.4.2.6 | Summary of Statistical Analysis of Plasma AX-158 Pharmacokinetic Data - Accumulation | PK Set |
| Figure 14.4.2.4 | Accumulation Least Squares Geometric Mean Ratios and 90% Cls of Plasma AX-158 Pharmacokinetic Data | PK Set |
| Table 14.4.2.7 | Summary of Urine AX-158 Concentration Data | PK Set |
| Table 14.4.2.8 | Summary of Derived Urine AX-158 Pharmacokinetic Data | PK Set |

## 14.5 Pharmacodynamics


Document Title:SAP Template - Phase 1Document Number:TEMP-00109Previous Document Number:STATt008



Not applicable.

#### 14.6 Other

Not applicable.

## **Subject Data: Listings Contained in Report Appendix 16.2**

16.2.1 Visit Dates, Dosing Information and Disposition

| Listing 16.2.1.1 | Visit Dates | Safety Set |
|------------------|---------------------------|----------------------|
| Listing 16.2.1.2 | Study Drug Administration | Safety Set |
| Listing 16.2.1.3 | Subject Disposition | All Consented<br>Set |
| Listing 16.2.1.4 | Additional Notes | Safety Set |

#### 16.2.2 Protocol Deviations

| Listing 16.2.2.1 Protocol Deviations | Safety Set |
|--------------------------------------|------------|
|--------------------------------------|------------|

### 16.2.3 Analysis Sets

| Listing 16.2.3.1 | Analysis Sets | All Randomised |
|------------------|---------------|----------------|
| | | Subjects |

## 16.2.4 Demographic Data and Other Baseline Characteristics

| Listing 16.2.4.1 | Demographic Information | Safety Set |
|------------------|-------------------------------------------|------------|
| Listing 16.2.4.2 | Substance Use History | Safety Set |
| Listing 16.2.4.3 | Medical History and Concurrent Conditions | Safety Set |
| Listing 16.2.4.4 | Virology Results | Safety Set |
| Listing 16.2.4.5 | COVID-19 Results | Safety Set |
| Listing 16.2.4.6 | Drugs of Abuse Results | Safety Set |
| Listing 16.2.4.7 | Inclusion/Exclusion Criteria Failures | Safety Set |

## 16.2.5 Drug Concentration Data and Pharmacokinetics

## 16.2.5 Drug Concentration Data and Pharmacokinetics

| Listing 16.2.5.1 | Plasma AX-158 Concentration Data | Safety Set |
|---|---|---|
| Figure 16.2.5.1 | Individual Plasma AX-158 Concentration-Time Curves on a Linear Scale | Safety Set |
| Figure 16.2.5.2 | Individual Plasma AX-158 Concentration-Time Curves on a Semi-Logarithmic Scale | Safety Set |

Version: 3.

Document Title:SAP Template - Phase 1Document Number:TEMP-00109Previous Document Number:STATt008





| Listing 16.2.5.2 | Individual Derived Plasma AX-158 Pharmacokinetic Parameters | Safety Set |
|---|---|---|
| Listing 16.2.5.3 | Raw Statistical Analysis of Plasma AX-158 Pharmacokinetic Data - Dose Proportionality | PK Set |
| Listing 16.2.5.4 | Raw Statistical Analysis of Plasma AX-158 Pharmacokinetic Data - Dose Independence | PK Set |
| Listing 16.2.5.5 | Raw Statistical Analysis of Plasma AX-158 Pharmacokinetic Data – Food Effect | PK Set |
| Listing 16.2.5.6 | Raw Statistical Analysis of Plasma AX-158 Pharmacokinetic Data - Steady State | PK Set |
| Listing 16.2.5.7 | Raw Statistical Analysis of Plasma AX-158 Pharmacokinetic Data - Accumulation | PK Set |
| Listing 16.2.5.8 | Urine AX-158 Concentration Data | PK Set |
| Listing 16.2.5.9 | Derived Urine AX-158 Pharmacokinetic Data | PK Set |

## 16.2.6 Efficacy

Not applicable.

Listing 16.2.7.1

#### 16.2.7 Adverse Events

Adverse Events

| 16.2.8 Individ | dual Laboratory Safety Measurements | |
|------------------|-------------------------------------|------------|
| Listing 16.2.8.1 | Biochemistry Data | Safety Set |
| Listing 16.2.8.2 | Hematology Data | Safety Set |
| Listing 16.2.8.3 | Coagulation Data | Safety Set |
| Listing 16.2.8.4 | Urinalysis Data | Safety Set |
| Listing 16.2.8.5 | Microscopy Data | Safety Set |
| Listing 16.2.8.6 | Other Laboratory Data | Safety Set |

### 16.2.9 Vital Signs

| Listing 16.2.9.1 | Vital Signs Data | Safety Set |
|------------------|------------------|------------|
|------------------|------------------|------------|

#### 16.2.10 Physical Examination

| Listing 16.2.10.1 | Physical Examination Data | Safety Set |
|-------------------|---------------------------|------------|
|-------------------|---------------------------|------------|

### 16.2.11 ECG

Listing 16.2.11.1 12-lead ECG Data Safety Set

### 16.2.12 Prior and Concomitant Medication


Document Title:SAP Template - Phase 1Document Number:TEMP-00109Previous Document Number:STATt008

Safety Set



Artax Biopharma Inc: AX-158-101 Statistical Analysis Plan Final v1.0 14DEC2022

Listing 16.2.12.1 Prior and Concomitant Medications

Safety Set

## 16.2.13 Pharmacodynamics

Not applicable.

#### 16.2.14 Other

Listing 16.2.14.1 PD Sampling

Safety Set



## 15 SHELLS FOR TABLES, FIGURES AND LISTINGS

The intended layouts for tables, figures and listings are presented. However, it may be appropriate to change the layouts, upon review of the data available, for completeness and clarity.

QCd output will be produced as Rich Text Format (.rtf) files for convenient inclusion in the CSR. The default tables, figures and listings (TFL) layout will be as follows:

| Orientation | A4 Landscape |
|---|---|
| Margins | Top: 2.54 cm Bottom: 2.54 cm Left: 2.54 cm Right: 2.54 cm |
| Font | Courier New 9pt |
| Headers<br>(Centre) | Sponsor Protocol Number, TFL Number, Title, Analysis Set |
| Footers<br>(Left) | Source Listing, Date/Time TFL Generated, Page Number, i.e. Page x of y |

Listing shells are displayed within this document without the comments field but, should there be any comments recorded for the represented data, this field will be added to the listing. In addition, at the time of programming, footnotes will be added to the listing, table or figure as needed. All footnotes will be used for purposes of clarifying the presentation.

Each table and figure will be produced for each study part (Part A, Part B or Part C) unless stated otherwise. The TFL title will include a suffix of ' – Part A' etc. Unless stated otherwise, listings will contain information from all study parts combined, with the exception of safety laboratory listings which will be created separately for each part due to file size.

Should the number of variables within a listing or table be too great to fit on one page without compromising clarity, then the variables will be split across multiple subsequent pages and key identifying variables replicated with these (i.e. subject number, visit etc). The differing pages will be identified using a sequential number which will follow the TFL title, i.e. xxxx - (1), xxxx - (2).

All final TFLs will be reported from SDTM and ADaM datasets. SDTM and ADaM details will be documented in a separate specification document.



AX-158-101
Table 14.1.1.1
Summary of Study Disposition - Part A (SAD)
All Consented Set

| | Placebo*<br>(Fasted)<br>(N=X) | Cohort 1: AX-158 5 mg (Fasted) (N=X) | Cohort 2: AX-158 10 mg (Fasted) (N=X) | Cohort 3: AX-158 15 mg (Fasted) (N=X) | Cohort 4: AX-158 25 mg (Fasted) (N=X) | Cohort 5: AX-158 50 mg (Fasted) (N=X) | AX-158<br>Overall<br>(N=X) | Overall<br>(N=X) |
|---|---|---|---|---|---|---|---|---|
| Consented <sup>[a]</sup> | | | | | | | | Х |
| Dosed | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Completed Study | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Study Termination | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Reason for Study Termination | | | | | | | | |
| ADVERSE EVENT | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| LOST TO FOLLOW-UP | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| WITHDRAWAL BY SUBJECT | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| STUDY TERMINATED BY SPONSOR | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| PHYSICIAN DECISION | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| PROTOCOL VIOLATION | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| DEATH | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| OTHER | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Safety Set | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| PK Set | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |

Source Listing: 16.2.1.2, 16.2.1.3, 16.2.3.1; Produced: yyyy-mm-ddThh:mm - Page x of y

Treatment: single dose of AX-158 capsule or placebo in the fasted state.

Percentages will be calculated from the number of dosed subjects within a treatment group.

[a] Subjects for whom Informed Consent was obtained, including screening failures/non-runners.


**Document Title:** SAP Template - Phase 1

<sup>\*</sup> Placebo subjects pooled across all cohorts.



## Artax Biopharma Inc: AX-158-101 Statistical Analysis Plan Final v1.0 14DEC2022

Programming Note: Additional SAD cohorts to be added as appropriate. A similar table will be produced for Part C (MAD) - 3 cohorts, where additional MAD cohorts can be added as appropriate, with the treatment footnote

• "Treatment: once daily dosing of AX-158 or placebo in a <fasted/fed> state for 10 days, with the final dose administered on the morning of Day 10.". This should be amended as appropriate if a once daily dosing regimen is not implemented.


**Document Title:** SAP Template - Phase 1



# AX-158-101 Table 14.1.1.1 Summary of Study Disposition - Part B (Food Effect) All Consented Set

| | Number of Subjects (%) |
|-------------------------------|------------------------|
| Consented | X |
| Screening Failure/Non-Runners | х |
| Dosed: | () |
| 15 mg AX-158 in fed state | x (x.x)<br>x (x.x) |
| 15 mg AX-158 in fasted state | |
| Completed Study | x (x.x) |
| Study Termination | x (x.x) |
| Reason for Study Termination | |
| ADVERSE EVENT | x (x.x) |
| LOST TO FOLLOW-UP | x (x.x) |
| WITHDRAWAL BY SUBJECT | x (x.x) |
| STUDY TERMINATED BY SPONSOR | x (x.x) |
| PHYSICIAN DECISION | x (x.x) |
| PROTOCOL VIOLATION | x (x.x) |
| DEATH | x (x.x) |
| OTHER | x (x.x) |
| Safety Set | x (x.x) |
| PK Set | x (x.x) |

Source Listing: 16.2.1.2, 16.2.1.3, 16.2.3.1; Produced: yyyy-mm-ddThh:mm - Page x of y
Treatment = a single dose of 15 mg AX-158 capsules over 2 treatment periods, in the fed and fasted state.
Percentages will be calculated from the number of dosed subjects within a treatment group.


**Document Title:** SAP Template - Phase 1



AX-158-101
Table 14.1.2.1
Summary of Demographic Information - Part A (SAD)
Safety Set

| Parameter | Statistic | Placebo*<br>(N=X) | Cohort 1: AX-158 5 mg (Fasted) (N=X) | | Cohort 5: AX-158 50 mg (Fasted) (N=X) | AX-158<br>Overall<br>(N=X) | Overall<br>(N=X) |
|---|---|---|---|---|---|---|---|
| Age (yrs) | n | X | x | X | X | X | X |
| Age (yis) | Mean | X.X | X . X | x.x | x.x | x.x | x.x |
| | SD | X.XX | X.XX | x.xx | X.XX | X.XX | X.XX |
| | Min | X | X | X | X | X | х |
| | Median | x.x | x.x | x.x | X.X | x.x | x.x |
| | Max | x | x | X | X | X | X |
| Height (m) | n | X | X | X | X | X | X |
| | Mean | X.X | X . X | x.x | X.X | x.x | x.x |
| | SD | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |
| | Min | X | X | X | Х | X | X |
| | Median | X . X | X . X | X.X | X.X | X.X | X.X |
| | Max | X | X | X | X | X | X |

Source Listing: 16.2.4.1; Produced: yyyy-mm-ddThh:mm - Page x of y

Treatment: single dose of AX-158 capsule or placebo in the fasted state.

Percentages calculated from the number of subjects in the Safety Set within a treatment group.

Programming Note: Similar tables will be presented for Part B (Food Effect) and Part C (MAD), with column headers and treatment footnotes as presented in Table 14.1.1.1.

[Continued overleaf...]


**Document Title:** SAP Template - Phase 1

<sup>\*</sup> Placebo subjects pooled across all cohorts.



AX-158-101
Table 14.1.2.1
Summary of Demographic Information - Part A (SAD)
Safety Set

| Parameter | Statistic | Placebo*<br>(N=X) | Cohort 1: AX-158 5 mg (Fasted) (N=X) | | Cohort 5: AX-158 50 mg (Fasted) (N=X) | AX-158<br>Overall<br>(N=X) | Overall<br>(N=X) |
|---|---|---|---|---|---|---|---|
| Weight (kg) | n | X | x | X | X | Х | Х |
| Weight (kg) | Mean | X . X | X.X | x.x | X.X | X.X | x.x |
| | SD | X.XX | X.XX | x.xx | X.XX | X.XX | x.xx |
| | Min | X | X | X | X | X | X |
| | Median | X • X | X • X | X • X | X.X | X.X | X.X |
| | Max | Х | X | Х | Х | X | X |
| BMI (kg/m²) | n | X | X | X | X | X | X |
| | Mean | X.X | X.X | x.x | X.X | x.x | x.x |
| | SD | X.XX | x.xx | X.XX | X.XX | X.XX | X.XX |
| | Min | X | X | X | Х | X | Х |
| | Median | X . X | X • X | X.X | X.X | X • X | X.X |
| | Max | X | X | X | X | X | X |

Source Listing: 16.2.4.1; Produced: yyyy-mm-ddThh:mm - Page x of y

Treatment: single dose of AX-158 capsule or placebo in the fasted state.

Percentages calculated from the number of subjects in the Safety Set within a treatment group.

Programming Note: Similar tables will be presented for Part B (Food Effect) and Part C (MAD), with column headers and treatment footnotes as presented in Table 14.1.1.1.

[Continued overleaf...]


**Document Title:** SAP Template - Phase 1

<sup>\*</sup> Placebo subjects pooled across all cohorts.





# AX-158-101 Table 14.1.2.1 Summary of Demographic Information - Part A (SAD) Safety Set

| Parameter | | Statistic | Placebo*<br>(N=X) | Cohort 1:<br>AX-158<br>5 mg<br>(Fasted)<br>(N=X) | | Cohort 5:<br>AX-158<br>50 mg<br>(Fasted)<br>(N=X) | AX-158<br>Overall<br>(N=X) | Overall (N=X) |
|---|---|---|---|---|---|---|---|---|
| Gender | MALE | n (%) | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) |
| | FEMALE | n (%) | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) |
| Ethnicity | NOT HISPANIC OR LATINO | n (%) | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) |
| | HISPANIC OR LATINO | n (%) | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) |
| Race | BLACK OR AFRICAN AMERICAN | n (%) | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) |
| | AMERICAN INDIAN OR ALASKA NATIVE | n (%) | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) |
| | ASIAN | n (%) | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) |
| | NATIVE HAWAIIAN OR OTHER PACIFIC ISLANDER | n (%) | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) |
| | WHITE | n (%) | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) |
| | MIXED | n (%) | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) |
| | OTHER | n (%) | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) |

Source Listing: 16.2.4.1; Produced: yyyy-mm-ddThh:mm - Page x of y

Treatment: single dose of AX-158 capsule or placebo in the fasted state.

Percentages calculated from the number of subjects in the Safety Set within a treatment group.

Programming Note: Similar tables will be presented for Part B (Food Effect) and Part C (MAD), with column headers and treatment footnotes as presented in Table 14.1.1.1.


**Document Title:** SAP Template - Phase 1

<sup>\*</sup> Placebo subjects pooled across all cohorts.



# AX-158-101 Table 14.3.1.1 Summary of Treatment Emergent Adverse Events - Part A (SAD) Safety Set

| | Placebo*<br>(N=X) | Cohort 1: AX-158 5 mg (Fasted) (N=X) | <br>AX-158<br>Overall<br>(N=X) | Overall<br>(N=X) |
|---|---|---|---|---|
| Number of TEAEs | x | Х | <br>Х | Х |
| Number (%) of subjects reporting at least | one: | | | |
| TEAE | x (x.x) | x (x.x) | <br>x (x.x) | x (x.x) |
| Serious TEAE | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| TEAE Leading to Withdrawal | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| TEAE Leading to Death | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Number (%) of subjects with TEAE by sever. | ity: | | | |
| MILD | x (x.x) | x (x.x) | <br>x (x.x) | x (x.x) |
| MODERATE | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| SEVERE | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Number (%) of subjects with TEAE by relat. | ionship | | | |
| to study drug: | | | | |
| REASONABLE POSSIBILITY | x (x.x) | x (x.x) | <br>x (x.x) | x (x.x) |
| NO REASONABLE POSSIBILITY | x (x.x) | x (x.x) | x (x.x) | x (x.x) |

Source Listing: 16.2.7.1; Produced: yyyy-mm-ddThh:mm - Page x of y

Treatment: single dose of AX-158 capsule or placebo in the fasted state.

A subject with multiple adverse events is counted only once at the maximum level of severity or the strongest relationship to treatment within each treatment category.

Percentages will be calculated from the number of subjects in the Safety Set within a treatment group.


**Document Title:** SAP Template - Phase 1

<sup>\*</sup> Placebo subjects pooled across all cohorts.



# AX-158-101 Table 14.3.1.1 Summary of Treatment Emergent Adverse Events - Part B (Food Effect) Safety Set

| | AX-158<br>15 mg<br>(Fasted)<br>(N=X) | AX-158<br>15 mg<br>(Fed)<br>(N=X) | Overall (N=X) |
|---|---|---|---|
| Number of TEAEs | х | Х | х |
| Number (%) of subjects reporting at least one | : | | |
| TEAE | x (x.x) | x (x.x) | x (x.x) |
| Serious TEAE | x (x.x) | x (x.x) | x (x.x) |
| TEAE Leading to Withdrawal | x (x.x) | x (x.x) | x (x.x) |
| TEAE Leading to Death | x (x.x) | x (x.x) | x (x.x) |
| Number (%) of subjects with TEAE by severity: | | | |
| MILD | x (x.x) | x (x.x) | x (x.x) |
| MODERATE | x (x.x) | x (x.x) | x (x.x) |
| SEVERE | x (x.x) | x (x.x) | x (x.x) |
| Number (%) of subjects with TEAE by relations to study drug: | hip | | |
| REASONABLE POSSIBILITY | x (x.x) | x (x.x) | x (x.x) |
| NO REASONABLE POSSIBILITY | x (x.x) | x (x.x) | x (x.x) |

Source Listing: 16.2.7.1; Produced: yyyy-mm-ddThh:mm - Page x of y

Treatment= a single dose of 15 mg AX-158 capsules over 2 treatment periods, in the fed and fasted state. A subject with multiple adverse events is counted only once at the maximum level of severity or the strongest relationship to treatment within each treatment category.

Percentages will be calculated from the number of subjects in the Safety Set within a treatment.


**Document Title:** SAP Template - Phase 1



## Artax Biopharma Inc: AX-158-101 Statistical Analysis Plan Final v1.0 14DEC2022

AX-158-101
Table 14.3.1.1
Summary of Treatment Emergent Adverse Events - Part C (MAD)
Safety Set

| | Placebo* <fed fasted="">) (N=X)</fed> | Cohort 1:<br>AX-158<br>5 mg<br>( <fed fasted="">)<br/>(N=X)</fed> | Cohort 2: AX-158 <x> mg (<fed fasted="">) (N=X)</fed></x> | Cohort 3:<br>AX-158<br><x> mg<br/>(<fed fasted="">)<br/>(N=X)</fed></x> | AX-158<br>Overall<br>(N=X) | Overall<br>(N=X) |
|---|---|---|---|---|---|---|
| Number of TEAEs | Х | Х | Х | Х | Х | X |
| Number (%) of subjects reporting at least one: | | | | | | |
| TEAE | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Serious TEAE | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| TEAE Leading to Withdrawal | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| TEAE Leading to Death | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Number (%) of subjects with TEAE by severity: | | | | | | |
| MILD | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| MODERATE | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| SEVERE | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| Number (%) of subjects with TEAE by relationship | | | | | | |
| to study drug: | | | | | | |
| REASONABLE POSSIBILITY | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| NO REASONABLE POSSIBILITY | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) | x (x.x) |

Source Listing: 16.2.7.1; Produced: yyyy-mm-ddThh:mm - Page x of y

Treatment: once daily dosing of AX-158 or placebo in a <fasted/fed> state for 10 days, with the final dose administered on the morning of Day 10.

A subject with multiple adverse events is counted only once at the maximum level of severity or the strongest relationship to treatment within each treatment category.

Percentages will be calculated from the number of subjects in the Safety Set within a treatment.

Programming Note: Treatment footnote should be amended as appropriate if a once daily dosing regimen is not implemented.

Version: 3.

**Document Title:** SAP Template - Phase 1

<sup>\*</sup> Placebo subjects pooled across all cohorts.



AX-158-101 Table 14.3.1.2

Summary of Treatment Emergent Adverse Events by System Organ Class and Preferred Term - Part A (SAD) Safety Set

| | | Number c | f Events | / Number (%) of | Subjects |
|---|---|---|---|---|---|
| | <del></del> | Cohort 1: | | | |
| | | AX-158 | | | |
| | | 5 mg | | AX-158 | |
| System Organ Class | Placebo* | (Fasted) | | Overall | Overall |
| Preferred Term | (N=X) | (N=X) | | (N=X) | (N=X) |
| CONCERN ODCAN CLASS | / /) | / () | | / () | / () |
| <system class="" organ=""></system> | x / x (x.x) | | • • • | x / x (x.x) | |
| <preferred term=""></preferred> | x / x (x.x) | x / x (x.x) | | x / x (x.x) | |
| <preferred term=""></preferred> | x / x (x.x) | x / x (x.x) | | x / x (x.x) | x / x (x.x) |
| <system class="" organ=""></system> | x / x (x.x) | x / x (x.x) | | x / x (x.x) | x / x (x.x) |
| <preferred term=""></preferred> | x / x (x.x) | x / x (x.x) | | x / x (x.x) | x / x (x.x) |

Source Listing: 16.2.7.1; Produced: yyyy-mm-ddThh:mm - Page x of y

Treatment: single dose of AX-158 capsule or placebo in the fasted state.

A subject is counted only once per SOC and PT within each treatment category.

Percentages will be calculated from the number of subjects in the Safety Set within a treatment group. MedDRA version 24.1.

Programming note: Similar tables will be presented for Part B (Food Effect) and Part C (MAD), with column headers and treatment footnotes as presented in Table 14.3.1.1.


**Document Title:** SAP Template - Phase 1

<sup>\*</sup> Placebo subjects pooled across all cohorts.



# AX-158-101 Table 14.3.1.3 Summary of Treatment Emergent Adverse Events by Preferred Term - Part A (SAD) Safety Set

| | | Number o | of Events | / Number (%) of | Subjects |
|---|---|---|---|---|---|
| | | Cohort 1: | | | |
| | | AX-158 | | | |
| | | 5 mg | | AX-158 | |
| | Placebo* | (Fasted) | | Overall | Overall |
| Preferred Term | (N=X) | (N=X) | | (N=X) | (N=X) |
| | , , , , | , , , | | , , , | , , , |
| <preferred term=""></preferred> | x / x (x.x) | x / x (x.x) | • • • | x / x (x.x) | |
| <preferred term=""></preferred> | x / x (x.x) | x / x (x.x) | | x / x (x.x) | x / x (x.x) |
| <preferred term=""></preferred> | x / x (x.x) | x / x (x.x) | | x / x (x.x) | x / x (x.x) |
| <preferred term=""></preferred> | | | | | |
| <preferred term=""></preferred> | x / x (x.x) | x / x (x.x) | | x / x (x.x) | x / x (x.x) |

Source Listing: 16.2.7.1; Produced: yyyy-mm-ddThh:mm - Page x of y

Treatment: single dose of AX-158 capsule or placebo in the fasted state.

A subject is counted only once per PT within each treatment category.

Percentages will be calculated from the number of subjects in the Safety Set within a treatment group. MedDRA version 24.1.

Programming Note: To be sorted in descending frequency of number of subjects in Overall column.

Programming note: Similar tables will be presented for Part B (Food Effect) and Part C (MAD), with column headers and treatment footnotes as presented in Table 14.3.1.1.


**Document Title:** SAP Template - Phase 1

<sup>\*</sup> Placebo subjects pooled across all cohorts.



AX-158-101 Table 14.3.1.4

Summary of Treatment Emergent Adverse Events by System Organ Class, Preferred Term and Severity - Part A (SAD)

Safety Set

| | | | Number | (%) of Su | bjects | |
|---|---|---|---|---|---|---|
| System Organ Class<br>Preferred Term | Severity | Placebo* | Cohort 1: AX-158 5 mg (Fasted) (N=X)) | | AX-158<br>Overall<br>(N=X) | Overall |
| <system class="" organ=""></system> | MILD | x (x.x) | x (x.x) | | x (x.x) | x (x.x) |
| | MODERATE | x (x.x) | x (x.x) | | x (x.x) | x (x.x) |
| | SEVERE | x (x.x) | x (x.x) | | x (x.x) | x (x.x) |
| <preferred term=""></preferred> | MILD | x (x.x) | x (x.x) | | x (x.x) | x (x.x) |
| <preferred term=""></preferred> | MILD | x (x.x) | x (x.x) | | x (x.x) | x (x.x) |
| <pre><pre><pre><pre><pre><pre><pre><pre></pre></pre></pre></pre></pre></pre></pre></pre> | MILD | x (x.x) | x (x.x) | | x (x.x) | x (x.x) |
| | MODERATE | x (x.x) | x (x.x) | | x (x.x) | x (x.x) |
| | SEVERE | x (x.x) | x (x.x) | | x (x.x) | x (x.x) |

Source Listing: 16.2.7.1; Produced: yyyy-mm-ddThh:mm - Page x of y

Treatment: single dose of AX-158 capsule or placebo in the fasted state.

A subject with multiple occurrences of an AE is counted only once at the maximum level of severity within a SOC, PT and treatment group.

Percentages will be calculated from the number of subjects in the Safety Set within a treatment group. MedDRA version 24.1.

Programming note: This table will be repeated for Similar tables will be presented for Part B (Food Effect) and Part C (MAD), with column headers and treatment footnotes as presented in Table 14.3.1.1.


**Document Title:** SAP Template - Phase 1

<sup>\*</sup> Placebo subjects pooled across all cohorts.



AX-158-101 Table 14.3.1.5

Summary of Treatment Emergent Adverse Events by System Organ Class, Preferred Term and Relationship - Part A (SAD)
Safety Set

| | | Number (%) of Subjects | | | |
|---|---|---|---|---|---|
| ystem Organ Class Preferred Term SYSTEM ORGAN CLASS TERM> <preferred term=""> <preferred term=""></preferred></preferred> | Relationship<br>to Study Drug | Placebo*<br>(N=X) | Cohort 1: AX-158 5 mg (Fasted) (N=X)) | AX-158<br>Overall<br>(N=X) | Overall<br>(N=X) |
| <system class="" organ="" term=""></system> | REASONABLE POSSIBILITY | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | NO REASONABLE POSSIBILITY | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| <preferred term=""></preferred> | REASONABLE POSSIBILITY | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| <preferred term=""></preferred> | REASONABLE POSSIBILITY | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| <preferred term=""></preferred> | NO REASONABLE POSSIBILITY | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| <preferred term=""></preferred> | REASONABLE POSSIBILITY | x (x.x) | x (x.x) | x (x.x) | x (x.x) |
| | NO REASONABLE POSSIBILITY | x (x.x) | x (x.x) | x (x.x) | x (x.x) |

Source Listing: 16.2.7.1; Produced: yyyy-mm-ddThh:mm - Page x of y

Treatment: single dose of AX-158 capsule or placebo in the fasted state.

A subject with multiple occurrences of an AE is counted only once at the strongest relationship to treatment within a SOC, PT and treatment group.

Percentages will be calculated from the number of subjects in the Safety Set within a treatment group. MedDRA version 24.1.

neabidi verbion 21.1.

Programming note: Similar tables will be presented for Part B (Food Effect) and Part C (MAD), with column headers and treatment footnotes as presented in Table 14.3.1.1.


**Document Title:** SAP Template - Phase 1

<sup>\*</sup> Placebo subjects pooled across all cohorts.



# AX-158-101 Table 14.3.1.6 Serious Adverse Events - Part A (SAD) - (1) Safety Set

<Treatment> OR <Cohort <X>: Treatment>

| | | System Organ Class/ | | | | | Time | |
|---|---|---|---|---|---|---|---|---|
| | Event | Preferred Term/ | Onset Date | End Date/ | Date | Duration | Post Dose | |
| Subject | Number | Reported Term | /Time | Time/Ongoing | Reported | (dd:hh:mm) | (dd:hh:mm) | Severity |
| | | , | | | | | | |
| XXX | X | xxxxxxxxx/ | XXXXXXX | XXXXXXX | XXXXXX | XX:XX:XX | XX:XX:XX | XXXXXXX |
| | | xxxxxxxx/ | Txx:xx | Txx:xx | | | | |
| | | XXXXXXXX | | | | | | |
| XXX | X | xxxxxxxx/ | xxxxxxx | XXXXXXX | xxxxxx | xx:xx:xx | xx:xx:xx | XXXXXXX |
| | | xxxxxxxxx/ | Txx:xx | Txx:xx | | | | |
| | | xxxxxxxx | | | | | | |
| | X | xxxxxxxx/ | XXXXXX | XXXXXX | XXXXXX | xx:xx:xx | xx:xx:xx | XXXXXXX |
| | | xxxxxxxxx/ | Txx:xx | Txx:xx | | | | |
| | | XXXXXXXX | | | | | | |
| XXX | Х | xxxxxxxxx/ | xxxxxxx | xxxxxxx | xxxxx | xx:xx:xx | xx:xx:xx | xxxxxxx |
| | | xxxxxxxx/ | Txx:xx | Txx:xx | | | | |
| | | xxxxxxxx | | | | | | |

Source Listing: 16.2.7.1; Produced: yyyy-mm-ddThh:mm - Page x of y Treatment: single dose of AX-158 capsule or placebo in the fasted state. SAE = Serious Adverse Event.

MedDRA version 24.1.

Programming note: Within a study part, AEs occurring prior to first dose of study drug and placebo AEs will be pooled across cohorts and presented first.

Programming Note: This table will be repeated for for Part B (Food Effect) and Part C (MAD), with treatment footnotes as presented in Table 14.3.1.1. Similar tables will be presented for Adverse Events Leading to Withdrawal - Parts A, B and C (Table 14.3.1.7) and Adverse Events Leading to Death - Parts A, B and C (Table 14.3.1.8).


**Document Title:** SAP Template - Phase 1



# AX-158-101 Table 14.3.1.6 Serious Adverse Events - Part A (SAD) - (2) Safety Set

<Treatment> OR <Cohort <X>: Treatment>

| Subject | Event<br>Number | System Organ Class/<br>Preferred Term/<br>Reported Term | Relationship<br>to Study Drug | SAE | SAE<br>Criteria | Action | Outcome | Comment |
|---|---|---|---|---|---|---|---|---|
| xxx | х | xxxxxxxx/<br>xxxxxxxxx/<br>xxxxxxxxx | xxxxxxx | х | xxxxxxxxxx | xxxxx | xxxxxx | xxxxxxxx |
| xxx | X | xxxxxxxx/<br>xxxxxxxxx/<br>xxxxxxxxx | xxxxxxx | Х | xxxxxxxxxx | xxxxx | xxxxxx | xxxxxxxx |
| | Х | xxxxxxxxx/<br>xxxxxxxxx/ | xxxxxxx | Х | xxxxxxxxxx | xxxxx | xxxxx | xxxxxxxx |
| xxx | х | xxxxxxxx/<br>xxxxxxxxx/<br>xxxxxxxxx | xxxxxxx | Х | xxxxxxxxxx | xxxxxx | xxxxxx | xxxxxxxx |

Source Listing: 16.2.7.1; Produced: yyyy-mm-ddThh:mm - Page x of y

Treatment: single dose of AX-158 capsule or placebo in the fasted state.

SAE = Serious Adverse Event.

MedDRA version 24.1.

Programming note: Within a study part, AEs occurring prior to first dose of study drug and placebo AEs will be pooled across cohorts and presented first.

Programming Note: This table will be repeated for for Part B (Food Effect) and Part C (MAD), with treatment footnotes as presented in Table 14.3.1.1. Similar tables will be presented for Adverse Events Leading to Withdrawal - Parts A, B and C (Table 14.3.1.7) and Adverse Events Leading to Death - Parts A, B and C (Table 14.3.1.8).


**Document Title:** SAP Template - Phase 1



# AX-158-101 Table 14.3.2.1 Biochemistry Out of Normal Range Data - Part A (SAD) Safety Set

<Treatment> OR <Cohort <X>: Treatment>

| | | | | | | | Norma | ıl Range | Alert Range | |
|---|---|---|---|---|---|---|---|---|---|---|
| Subject | Visit/<br>Time Point | Sample<br>Date/Time | Sample<br>ID | Parameter<br>(Unit) | Result | Flag | Low | High | Low | High |
| XXX | XXXXXX | XXXXXXXXX | XXXXX | XXXXXXX | X.XX | X | X.X | X.XX | X.X | X.XX |
| | | | | XXXXXXX | X.XX | X | X.X | X.XX | X.X | X.XX |
| | | | | XXXXXXX | X.XX | X | X.X | X.XX | X.X | X.XX |
| | | | | XXXXXXX | X.XX | X | X . X | X.XX | X . X | X.XX |
| | | | | xxxxxx | x.xx | X | X.X | x.xx | X.X | X.XX |
| | xxxxxx | xxxxxxxxx | xxxxx | xxxxxx | X.XX | x | x.x | X.XX | X • X | X.XX |
| | | | | XXXXXXX | X.XX | X | X . X | X.XX | X . X | X.XX |
| | | | | XXXXXXX | X.XX | X | X.X | X.XX | X.X | X.XX |
| | | | | XXXXXX | X.XX | X | X.X | X.XX | X . X | X.XX |
| | | | | XXXXXXX | X.XX | X | X.X | X.XX | X.X | X.XX |

Source Listing: 16.2.8.1; Produced: yyyy-mm-ddThh:mm - Page x of y

Treatment: single dose of AX-158 capsule or placebo in the fasted state.

H\* = Above Alert Range; H = Above Normal Range; Lo = Below Normal Range; L\* = Below Alert Range.

Programming Note: This table will be repeated for for Part C (MAD), with treatment footnote as presented in Table 14.1.1.1. Similar tables will be produced for Hematology Out of Normal Range Data - Parts A and C (Table 14.3.2.2), Coagulation Out of Normal Range Data - Parts A and C (Table 14.3.2.3) and Urinalysis Out of Normal Range Data - Parts A and C (Table 14.3.2.4 - no alert ranges for urinalysis).


**Document Title:** SAP Template - Phase 1



AX-158-101
Table 14.3.2.1
Biochemistry Out of Normal Range Data - Part B (Food Effect)
Safety Set

| | | | | | | | | | Norma | l Range | Aler | t Range |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject | Study<br>Period | Treatment | Visit | Sample<br>Date/Time | Sample<br>ID | Parameter<br>(Unit) | Result | Flag | Low | High | Low | High |
| XXX | X | XXXXXXX | XXXX | XXXXXXXXX | XXXXX | XXXXXXX | X.XX | X | X.X | X.XX | X.X | X.XX |
| | | | | | | XXXXXXX | X.XX | X | X.X | X.XX | X.X | X.XX |
| | | | | | | XXXXXXX | X.XX | X | X.X | X.XX | X.X | X.XX |
| | | | | | | XXXXXXX | X.XX | X | X . X | X.XX | X.X | X.XX |
| | | | | | | xxxxxx | X.XX | X | X.X | X.XX | X.X | X.XX |
| | Х | xxxxxxx | XXXX | xxxxxxxxx | XXXXX | xxxxxx | X.XX | Х | x.x | X.XX | x.x | x.xx |
| | | | | | | XXXXXXX | X.XX | X | X . X | X.XX | X.X | X.XX |
| | | | | | | XXXXXXX | X.XX | X | X . X | X.XX | X.X | X.XX |
| | | | | | | XXXXXXX | X.XX | X | X . X | X.XX | X.X | X.XX |
| | | | | | | XXXXXXX | X.XX | X | X.X | X.XX | X.X | x.xx |

Source Listing: 16.2.8.1; Produced: yyyy-mm-ddThh:mm - Page x of y Treatment= a single dose of 15 mg AX-158 capsules over 2 treatment periods, in the fed and fasted state.

H\* = Above Alert Range; H = Above Normal Range; Lo = Below Normal Range; L\* = Below Alert Range.

Programming Note: Similar tables will be produced for Hematology Out of Normal Range Data - Part B (Table 14.3.2.2), Coagulation Out of Normal Range Data - Part B (Table 14.3.2.3) and Urinalysis Out of Normal Range Data - Part B (Table 14.3.2.4 - no alert ranges for urinalysis).


**Document Title:** SAP Template - Phase 1



AX-158-101 Table 14.3.2.5

Summary of Absolute and Change from Baseline Biochemistry Results - Part A (SAD) Safety Set

#### <Parameter (<units>)>

| isit/<br>ime Point | n | Mean | SD | Min | Median | ., | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | median | Max | n | Mean | SD | Min | Median | Max |
| VISIT> | Х | x.xx | x.xxx | х.х | x.xx | X.X | | | | | | |
| VISIT> | X | X.XX | X.XXX | X.X | X.XX | X . X | | | | | | |
| VISIT> | X | X.XX | X.XXX | X.X | X.XX | X.X | | | | | | |
| VISIT> | X | X.XX | X.XXX | X.X | X.XX | X.X | Х | X.XX | X.XXX | X.X | X.XX | X.X |
| VISIT> | Х | X.XX | X.XXX | X . X | X.XX | X . X | Х | X.XX | X.XXX | x.x | x.xx | X.X |
| VISIT> | Х | X.XX | X.XXX | X.X | X.XX | X . X | Х | X.XX | X.XXX | x.x | x.xx | X.X |
| ファファフ | ISIT><br>ISIT><br>ISIT><br>ISIT> | X | X | ISIT> x x.xx x.xx ISIT> x x.xx x.xx ISIT> x x.xx x.xx ISIT> x x.xx x.xx | ISIT> x x.xx x.xx x.xx ISIT> x x.xx x.xx x.xx ISIT> x x.xx x.xx x.xx ISIT> x x.xx x.xx x.xx | ISIT> X X.XX X.XX X.XX ISIT> X X.XX X.XX X.XX ISIT> X X.XX X.XX X.XX ISIT> X X.XX X.XX X.XX | ISIT> X X.XX < | ISIT> X X.XX < | ISIT> X X.XX < | ISIT> X X.XX X.XXX X.XX X.XX | ISIT> X X.XX < | ISIT> |

Source Listing: Listing 16.2.8.1; Produced: yyyy-mm-ddThh:mm - Page x of y Treatment: single dose of AX-158 capsule or placebo in the fasted state. Baseline defined per subject as the last available assessment prior to dosing.

Programming Note: This table will be repeated for Part B and Part C, with visit/time points as appropriate and treatment footnotes as per Table 14.1.1.1. Similar tables will be produced for Summary of Absolute and Change from Baseline Hematology Results - Parts A, B and C (Table 14.3.2.6) and Summary of Absolute and Change from Baseline Coagulation Results - Parts A, B and C (Table 14.3.2.7).


**Document Title:** SAP Template - Phase 1

**Document Number:** TEMP-00109 **Previous Document Number:** STATt008



AX-158-101 Table 14.3.3.1

Summary of Absolute and Change from Baseline Vital Signs Data - Part A (SAD)
Safety Set

#### <Parameter (<units>)>

| | | | | Abso | olute | | | | Ch | ange f | rom B | aseline | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment | Visit/<br>Time Point | n | Mean | SD | Min | Median | Max | n | Mean | SD | Min | Median | Max |
| Placebo / | $<\!\!VISIT\!\!>$ | X | X.X | X.XX | X | X . X | X | | | | | | |
| Cohort <x>:</x> | $<\!\!VISIT\!\!>$ | X | X.X | X.XX | X | X . X | X | | | | | | |
| <x> mg AX-158</x> | $<\!\!\mathit{VISIT}\!\!>$ | X | X.X | X.XX | X | X . X | X | | | | | | |
| (Fasted) | $<\!\!\mathit{VISIT}\!\!>$ | Х | X.X | X.XX | Х | X . X | X | Х | X.X | X.XX | X | X . X | X |
| , | $<\!\!\!\!\!\!\!\!\!\!\!\!\!\!\!\!\!\!\!\!\!\!\!\!\!\!\!\!\!\!\!\!\!\!\!\!$ | X | X.X | X.XX | Х | X.X | X | Х | X.X | x.xx | X | X . X | Х |
| (N=x) | $<\!\!\!\!\!\!\!\!\!\!\!\!\!\!\!\!\!\!\!\!\!\!\!\!\!\!\!\!\!\!\!\!\!\!\!\!$ | X | X.X | X.XX | Х | X.X | X | Х | X.X | x.xx | X | X . X | Х |
| | $<\!\!VISIT\!\!>$ | Х | X.X | X.XX | Х | X.X | X | Х | X.X | x.xx | Х | X . X | Х |
| | $<\!\!VISIT\!\!>$ | Х | X.X | X.XX | Х | X.X | X | Х | X.X | x.xx | Х | X . X | Х |
| | $<\!\!\mathit{VISIT}\!\!>$ | X | X.X | X.XX | X | X.X | X | Х | X.X | x.xx | Х | X . X | X |
| | $<\!\!\!\!\!\!\!\!\!\!\!\!\!\!\!\!\!\!\!\!\!\!\!\!\!\!\!\!\!\!\!\!\!\!\!\!$ | X | X.X | X.XX | Х | X.X | Х | Х | X.X | x.xx | Х | X . X | Х |
| | $<\!\!VISIT\!\!>$ | Х | X.X | X.XX | Х | X.X | X | Х | X.X | x.xx | Х | X . X | Х |
| | <visit></visit> | Х | X . X | X.XX | Х | X.X | X | Х | Х.Х | X.XX | Х | X.X | Х |

Source Listing: 16.2.9.1; Produced: yyyy-mm-ddThh:mm - Page x of y

Treatment: single dose of AX-158 capsule or placebo in the fasted state.

Baseline defined per subject as the last available pre-dose result at each treatment period.

Programming Note: This table will be repeated for Part B and Part C, with visit/time points as appropriate and treatment footnotes as per Table 14.1.1.1.


**Document Title:** SAP Template - Phase 1



AX-158-101 Table 14.3.4.1

Summary of Absolute and Change from Baseline 12-Lead ECG Data - Part A (SAD) Safety Set

#### <Parameter (<units>)>

| | | | Absc | lute | | | Change from Baseline | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit/<br>Time Point | n | Mean | SD | Min | Median | Max | n | Mean | SD | Min | Median | Max |
| <visit></visit> | Х | x.x | x.xx | Х | x.x | X | | | | | | |
| <visit></visit> | Х | X.X | x.xx | Х | X • X | Х | | | | | | |
| <visit></visit> | Х | X . X | X.XX | Х | X . X | Х | | | | | | |
| < <i>VISIT</i> > | Х | X.X | X.XX | Х | X • X | Х | Х | X.X | x.xx | Х | X . X | Х |
| <visit></visit> | Х | X.X | X.XX | Х | X.X | Х | Х | X.X | X.XX | Х | X.X | Х |
| $<\!\!\mathit{VISIT}\!\!>$ | Х | X.X | X.XX | Х | X.X | Х | Х | X.X | x.xx | Х | X.X | Х |
| $<\!\!\mathit{VISIT}\!\!>$ | Х | X.X | X.XX | Х | X.X | X | Х | X.X | X.XX | Х | X.X | X |
| $<\!\!\mathit{VISIT}\!\!>$ | Х | X . X | X.XX | Х | X . X | X | Х | X.X | X.XX | X | X . X | X |
| $<\!\!\mathit{VISIT}\!\!>$ | Х | X . X | X.XX | X | X . X | X | Х | X.X | X.XX | X | X . X | X |
| | Time Point <visit> <visit></visit></visit></visit></visit></visit></visit></visit></visit></visit></visit></visit> | Time Point n | Time Point n Mean Color | Visit/<br>Time Point n Mean SD <visit> x x.x x.xx <visit> x x.x x.xx</visit></visit></visit></visit></visit></visit></visit></visit> | Time Point n Mean SD Min SD Min SD | Visit/<br>Time Point n Mean SD Min Median <visit> x x.x x.xx x.x <visit> x x.x x.xx x.x</visit></visit></visit></visit></visit></visit></visit> | Visit/<br>Time Point n Mean SD Min Median Max <visit> x x.x x.xx x.x x.x</visit> | Visit/<br>Time Point n Mean SD Min Median Max n <visit> x x.x x.xx x.x x.x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x<!--</td--><td>Visit/<br/>Time Point n Mean SD Min Median Max n Mean <visit> x x.x x.xx x.x x.x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x</visit></td><td>Visit/<br/>Time Point Nean SD Min Median Max n Mean SD <visit> x x.x x.xx x x.x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x</visit></td><td>Visit/<br/>Time Point Nean SD Min Median Max Nean SD Min <visit> X X.X X.XX X.X X.X X.X X.X X.X X.X X.X X.X X.X X.X X.X X.X X.X X.X X.X X.X X.X X.X X.X X.X X.X X.X X.X X.X X.X X.X X.X X.X X.X X.X X.X X.X X.X X.X X.X X.X X.X X.X X.X X.X X.X X.X X.X X.X X.X X.X X.X X.X X.X X.X X.X X.X X.X X.X X.X X.X X.X X.X X.X X.X X.X X.X X.X X.X X.X X.X X.X X.X X.X X.X X.X X.X X.X X.X X.X X.X X.X X.X X.X X.X X.X X.X</visit></td><td>Visit/ Time Point n Mean SD Min Median Max n Mean SD Min Median</td></visit> | Visit/<br>Time Point n Mean SD Min Median Max n Mean <visit> x x.x x.xx x.x x.x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x</visit> | Visit/<br>Time Point Nean SD Min Median Max n Mean SD <visit> x x.x x.xx x x.x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x</visit> | Visit/<br>Time Point Nean SD Min Median Max Nean SD Min <visit> X X.X X.XX X.X X.X</visit> | Visit/ Time Point n Mean SD Min Median Max n Mean SD Min Median |

Source Listing: 16.2.11.1; Produced: yyyy-mm-ddThh:mm - Page x of y

Treatment: single dose of AX-158 capsule or placebo in the fasted state.

Baseline defined per subject as the last available assessment prior to dosing.

Programming Note: This table will be repeated for Part B and Part C, with visit/time points as appropriate and treatment footnotes as per Table 14.1.1.1.


**Document Title:** SAP Template - Phase 1





AX-158-101
Table 14.3.4.2
Summary of 12-Lead ECG QTcF Categories - Part A (SAD)
Safety Set

| | | | Number of Subjects (%) | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment | Visit/Time<br>Point | ~ | TcF<=<br>0 mSec | | <= QTcF<br>80 mSec | | <= QTcF | ~ | TcF ><br>0 mSec | Dec | QTcF<br>reased/<br>Change | In | QTcF<br>crease<br>30 mSec | In | < QTcF<br>crease<br>50 mSec | In | QTcF<br>crease<br>0 mSec |
| Dlacaba / | <visit></visit> | Х | (x.x) | Х | , , | Х | (x.x) | Х | (x.x) | | | | | | | | |
| Placebo / | $<\!\!\mathit{VISIT}\!\!>$ | X | (x.x) | X | (x.x) | X | (x.x) | Х | (x.x) | | | | | | | | |
| Cohort <x>:</x> | $<\!\!VISIT\!\!>$ | X | (x.x) | X | (x.x) | X | (x.x) | X | (x.x) | X | (x.x) | X | (x.x) | X | (x.x) | X | (x.x) |
| $\langle X \rangle$ mg AX-158 | $<\!\!VISIT\!\!>$ | X | (x.x) | X | (x.x) | X | (x.x) | Х | (x.x) | X | (x.x) | X | (x.x) | X | (x.x) | X | (x.x) |
| (Fasted) | $<\!\!VISIT\!\!>$ | X | (x.x) | Х | (x.x) | X | (x.x) | Х | (x.x) | Х | (x.x) | X | (x.x) | Х | (x.x) | Х | (x.x) |
| (N=x) | $<\!\!VISIT\!\!>$ | Х | (x.x) | Х | (x.x) | Х | (x.x) | Х | (x.x) | Х | (x.x) | X | (x.x) | Х | (x.x) | Х | (x.x) |
| (11 21) | $<\!\!VISIT\!\!>$ | Х | (x.x) | Х | (x.x) | Х | (x.x) | Х | (x.x) | Х | (x.x) | Х | (x.x) | Х | (x.x) | Х | (x.x) |
| | <visit></visit> | Х | (x.x) | Х | (x.x) | х | (x.x) | Х | (x.x) | Х | (x.x) | Х | (x.x) | Х | (x.x) | Х | (x.x) |
| | <visit></visit> | Х | (x.x) | Х | (x.x) | х | (x.x) | Х | (x.x) | Х | (x.x) | Х | (x.x) | Х | (x.x) | Х | (x.x) |
| | <visit></visit> | Х | (x.x) | Х | (x.x) | х | (x.x) | Х | (x.x) | Х | (x.x) | Х | (x.x) | Х | (x.x) | Х | (x.x) |
| | <visit></visit> | Х | (x.x) | х | (x.x) | х | (x.x) | х | (x.x) | Х | (x.x) | х | (x.x) | х | (x.x) | Х | (x.x) |
| | <visit></visit> | Х | (x.x) | Х | (x.x) | Х | (x.x) | Х | (x.x) | Х | (x.x) | Х | (x.x) | Х | (x.x) | Х | (x.x) |

Source Listing: Listing 16.2.11.1; Produced: yyyy-mm-ddThh:mm; Page x of y Treatment: single dose of AX-158 capsule or placebo in the fasted state. Baseline defined per subject as the last available assessment prior to dosing. Percentages calculated from the number of non-missing observations.

Programming Note: This table will be repeated for Part B and Part C, with visit/time points as appropriate and treatment footnotes as per Table 14.1.1.1.


**Document Title:** SAP Template - Phase 1



 $\begin{array}{c} {\rm AX-158-101} \\ {\rm Table} \ 14.4.1.1 \\ {\rm Summary} \ {\rm of} \ {\rm Plasma} \ {\rm AX-158} \ {\rm Concentration} \ {\rm Data} \ - \ {\rm Part} \ {\rm A} \ ({\rm SAD}) \\ {\rm PK} \ {\rm Set} \end{array}$ 

| | | AX-158 Concentration ( <units>)</units> | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | Visit/ | | | Geometri | .C | | | | |
| Treatment | Time Point | n | Mean | Mean | SD | %CV | Minimum | Median | Maximum |
| Placebo / Cohort <x>:</x> | <visit>/<time point=""> <visit>/<time point=""></time></visit></time></visit> | X<br>X | x.xx<br>x.xx | X.XX<br>X.XX | x.xxx<br>x.xxx | x.x<br>x.x | X.X<br>X.X | X.XX<br>X.XX | X.X<br>X.X |
| <x> mg AX-158<br/>(Fasted)<br/>(N=x)</x> | <pre><visit>/<time point=""> <visit>/<time point=""></time></visit></time></visit></time></visit></time></visit></time></visit></time></visit></time></visit></time></visit></time></visit></time></visit></time></visit></time></visit></pre> | x<br>x<br>x<br>x<br>x<br>x<br>x | x.xx<br>x.xx<br>x.xx<br>x.xx<br>x.xx<br>x.xx<br>x.xx<br>x.x | x.xx<br>x.xx<br>x.xx<br>x.xx<br>x.xx<br>x.xx<br>x.xx<br>x.x | x.xx<br>x.xx<br>x.xxx<br>x.xxx<br>x.xxx<br>x.xxx<br>x.xxx<br>x.xxx | x.x | x.x | x.xx<br>x.xx<br>x.xx<br>x.xx<br>x.xx<br>x.xx<br>x.xx<br>x.x | x.x |
| | <visit>/<time point=""><br/><visit>/<time point=""></time></visit></time></visit> | X<br>X | x.xx<br>x.xx | x.xx<br>x.xx | X.XXX<br>X.XXX | x.x<br>x.x | x.x<br>x.x | x.xx<br>x.xx | X.X<br>X.X |

Source Listing: 16.2.5.1; Produced: yyyy-mm-ddThh:mm - Page x of y Treatment: single dose of AX-158 capsule or placebo in the fasted state.

Lower Limit of Quantitation – xx.xx < units. BLQ values set to 0 at pre-dose and LLOQ/2 for post-dose samples. In order to capture the zero values within the calculation of the geometric mean, a value of 0.001 was added to all pre-dose values prior to log-transformation. The geometric means were then calculated and 0.001 subtracted from the estimate, i.e. geometric mean = exp(mean of log(concentration+0.001)) - 0.001.

Programming note: This table will be repeated for Part B and Part C, with visit/time points as appropriate and treatment footnotes as per Table 14.1.1.1.


**Document Title:** SAP Template - Phase 1



#### AX-158-101 Figure 14.4.1.1

Geometric Mean Plasma AX-158 Concentration-Time Curves on a Linear Scale - Part A (SAD)

PK Set

```
Figure Specifications

By: Treatment, with all treatments on one plot

x axis: Time
x axis: Label: Time (h)
x axis: values: Day 1, Pre-dose, 30 min, 45 min, 1h, 2h, 3h, 4h, 6h, 8h, 12h, 24h, 36h, 48h, 72h (x-axis should present sampling time points only)

Y axis: Geometric mean concentration
Y axis Label: Geo. Mean AX-158 Conc. (<units>)
Y axis values: As appropriate

Legend (different line style/colour/symbol for each treatment):

Cohort <X>: AX-158 <X> mg (Fasted) (N=X)
```

Source Listing: 16.2.5.1; Produced: yyyy-mm-ddThh:mm - Page x of y Treatment: single dose of AX-158 capsule or placebo in the fasted state.

Lower Limit of Quantification = xx.xx < units >. BLQ values set to zero at pre-dose and LLOQ/2 for post-dose samples.

In order to capture the zero values within the calculation of the geometric mean, a value of 0.001 was added to all pre-dose values prior to log-transformation. The geometric means were then calculated and 0.001 subtracted from the estimate, i.e.  $\frac{1}{1000}$  geometric mean =  $\frac{1}{1000}$  exp (mean of log(concentration+0.001)) - 0.001.

Programming note: This figure will be repeated for Part B (Food Effect) and Part C by Day (MAD), with treatment footnotes as per Table 14.1.1.1. Similar figures will be produced for Geometric Mean Plasma AX-158 Concentration-Time Curves on a Semi-Logarithmic Scale (Figure 14.4.1.2).


**Document Title:** SAP Template - Phase 1



## Artax Biopharma Inc: AX-158-101 Statistical Analysis Plan Final v1.0 14DEC2022

AX-158-101 Table 14.4.2.1

Summary of Derived Plasma AX-158 Pharmacokinetic Parameters - Part A (SAD)  $$\operatorname{PK}$$  Set

| Treatment | Summary<br>Statistic | C <sub>max</sub><br>( <units>)</units> | $T_{max}$ ( <units>)</units> | AUC <sub>0-t</sub><br>( <units>)</units> | AUC <sub>0-24</sub> ( <units>)</units> | AUC <sub>0-inf</sub> ( <units>)</units> | AUC <sub>%extrap</sub> ( <units>)</units> | t <sub>1/2</sub><br>( <units>)</units> | $\lambda_z$ (1/h) | CL/F<br>( <units>)</units> | Vz/F<br>( <units>)</units> |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Cohort <x>:</x> | n | X | X | X | X | X | X | X | X | X | X |
| AX-158 < X > mg | Mean | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |
| (N=x) | Geo. Mean | X.XX | N/A | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |
| | SD | X.XXX | X.XXX | X.XXX | X.XXX | X.XXX | X.XXX | X.XXX | X.XXX | X.XXX | X.XXX |
| | CV% | X . X | X . X | X . X | X . X | X . X | X . X | X . X | X . X | X . X | X . X |
| | Min | X . X | X . X | X . X | X . X | X . X | X.X | X.X | X.X | X . X | X . X |
| | Median | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |
| | Max | X.X | X.X | X.X | x.x | X.X | x.x | x.x | X.X | X.X | X.X |

Source Listing: 16.2.5.2; Produced: yyyy-mm-ddThh:mm - Page x of y

Treatment: single dose of AX-158 capsule or placebo in the fasted state.

Lower Limit of Quantification = xx.xx < units >. For the purposes of PK parameter calculation, BLQ values were set to zero at predose and missing for post-dose time points.

N/A = Not applicable.

Programming note: This table will be repeated for Part B (Food Effect) and Part C (MAD) (for Day 1 and Day 10), with treatment footnotes as per Table 14.1.1.1.

Programming note: A similar table will be presented for Table 14.4.2.8 Summary of Derived Urine AX-158 Pharmacokinetic Data.


**Document Title:** SAP Template - Phase 1



 $\begin{array}{c} {\rm AX-158-101} \\ {\rm Table~14.4.2.2} \\ {\rm Summary~of~Statistical~Analysis~of~Plasma~AX-158~Dose~Proportionality~-~Part~A~(SAD)} \\ {\rm PK~Set} \end{array}$ 

| | | Geometric LSMear | ns (95% CI) | | | |
|---|---|---|---|---|---|---|
| _ | Cohort 1:<br>AX-158<br>5 mg | Cohort 2:<br>AX-158<br>10 mg | | Cohort 5:<br>AX-158<br>50 mg | _ | |
| Parameter | (N=X) | (N=X) | • • • | (N=X) | Intercept | Slope (95% CI) |
| C <sub>max</sub> ( <units>)</units> | x.xx<br>(x.xx, x.xx) | x.xx<br>(x.xx, x.xx) | | x.xx<br>(x.xx, x.xx) | x.xxx | x.xxx (x.xxx, x.xxx) |
| AUC <sub>0-t</sub> ( <units>)</units> | x.xx<br>(x.xx, x.xx) | x.xx<br>(x.xx, x.xx) | | x.xx<br>(x.xx, x.xx) | x.xxx | x.xxx (x.xxx, x.xxx) |
| AUC <sub>0-inf</sub> ( <units>)</units> | x.xx<br>(x.xx, x.xx) | x.xx<br>(x.xx, x.xx) | | x.xx<br>(x.xx, x.xx) | x.xxx | x.xxx (x.xxx, x.xxx) |
| AUC <sub>0-24</sub> ( <units>)</units> | x.xx<br>(x.xx, x.xx) | x.xx<br>(x.xx, x.xx) | ••• | x.xx<br>(x.xx, x.xx) | x.xxx | x.xxx (x.xxx, x.xxx) |

Source Listing: 16.2.5.2; Produced: yyyy-mm-ddThh:mm Page x of y

Treatment: single dose of AX-158 capsule or placebo in the fasted state.

Results obtained using a regression analysis on log-transformed values versus log-transformed dose using the power model.

Programming Note: A similar table will be presented for Part C (MAD), including  $C_{\text{max}}$  and  $AUC_{0-\text{tau}}$  results for Day 1 and Day 10 and  $AUC_{0-\text{inf}}$  results for Day 10, with treatment footnote as presented in Table 14.3.1.1.


**Document Title:** SAP Template - Phase 1



AX-158-101
Table 14.4.2.3
Summary of Statistical Analysis of Plasma AX-158 Dose Independence - Part A (SAD)
PK Set

| | | LSMeans (9 | 5% CI) | | | |
|---|---|---|---|---|---|---|
| Parameter | Cohort 1:<br>AX-158<br>5 mg<br>(N=X) | Cohort 2:<br>AX-158<br>10 mg<br>(N=X) | | Cohort 5:<br>AX-158<br>50 mg<br>(N=X) | Intercept | Slope (95% C.I.) |
| t <sub>1/2</sub> ( <units>)</units> | x.xx<br>(x.xx, x.xx) | x.xx<br>(x.xx, x.xx) | | | x.xxx | x.xxx (x.xxx, x.xxx) |
| CL/F ( <units>)</units> | x.xx<br>(x.xx, x.xx) | x.xx<br>(x.xx, x.xx) | | | x.xxx | x.xxx (x.xxx, x.xxx) |

Source Listing: 16.2.5.2; Produced: yyyy-mm-ddThh:mm - Page x of y

Treatment: single dose of AX-158 capsule or placebo in the fasted state.

Results obtained using a fixed effects ANOVA on non-transformed data with a fixed effect of dose.

Programming Note: A similar table will be presented for Part C (MAD), including results for final dosing day (Day 10), with treatment footnote as presented in Table 14.3.1.1.


**Document Title:** SAP Template - Phase 1



AX-158-101 Figure 14.4.2.1

Dose Response of Derived Plasma AX-158 Pharmacokinetic Parameters - Part A (SAD)  $_{\mbox{\footnotesize{PK}}}$  Set

< parameter (<units>) >

#### Figure Specifications

Procedure: SGPLOT

By: Parameter, one parameter per page

x axis: Dose

x axis: Label: AX-158 Dose (mg)
x axis: values: All dose levels

Y axis Geometric LSMeans and 95% CI for  $C_{max}$ ,  $AUC_{0-t}$  and  $AUC_{0-inf}$ ; LSMeans and 95% CI for and  $t_{1/2}$  and CL/F - overlaid with individual subject

values

Y axis Label: Geo. LSMeans (95% CI) for  $C_{\text{max}}\,,\,\text{AUC}_{0\text{-t}}\,\,\text{and}\,\,\text{AUC}_{0\text{-inf}}$ 

LSMeans (95% CI) for and  $t_{1/2}$  and CL/F

Y axis values: As Appropriate

Legend: Not Applicable

Source Listing: 16.2.5.2; Produced: yyyy-mm-ddThh:mm Page x of y

Treatment: single dose of AX-158 capsule or placebo in the fasted state.

Results for  $C_{\text{max}}$ ,  $AUC_{0-t}$  and  $AUC_{0-inf}$  obtained using a regression analysis on log-transformed values versus log-transformed dose using the power model. Results for CL/F and  $t_{1/2}$  obtained using a fixed effects ANOVA on non-transformed data with a fixed effect of dose.

Programming Note: A similar figure will be presented for Part C (MAD), including  $C_{\text{max}}$  and  $AUC_{0-\text{tau}}$  results for Day 1 and Day 10 and  $AUC_{0-\text{inf}}$ ,  $t_{1/2}$  and CL/F for Day 10, with treatment footnote as presented in Table 14.3.1.1.


**Document Title:** SAP Template - Phase 1





# $\begin{array}{c} {\rm AX-158-101} \\ {\rm Table} \ 14.4.2.4 \\ {\rm Summary} \ {\rm of} \ {\rm Statistical} \ {\rm Analysis} \ {\rm of} \ {\rm Plasma} \ {\rm AX-158} \ {\rm Food} \ {\rm Effect} \ - \ {\rm Part} \ {\rm B} \\ {\rm PK} \ {\rm Set} \end{array}$

| | Geometric LSN | Means (95% CI) | Geometric LSMean Ratio (%)<br>(90% CI)<br>[Within-Subject CV%] |
|---|---|---|---|
| Parameter | 15 mg AX-158<br>- Fed<br>(N=x) | 15 mg AX-158<br>- Fasted<br>(N=x) | Fed / Fasted |
| C <sub>max</sub> ( <units>)</units> | xx.x<br>(xx.x - xx.x) | xx.x<br>(xx.x - xx.x) | xx.x<br>(xx.x - xx.x)<br>[xx.x] |
| AUC <sub>0-t</sub> ( <units>)</units> | xx.x<br>(xx.x - xx.x) | xx.x<br>(xx.x - xx.x) | xx.x<br>(xx.x - xx.x)<br>[xx.x] |
| AUC <sub>0-inf</sub> ( <units>)</units> | xx.x<br>(xx.x - xx.x) | xx.x<br>(xx.x - xx.x) | xx.x<br>(xx.x - xx.x)<br>[xx.x] |

Source Listing: 16.2.5.2 Produced: yyyy-mm-ddThh:mm - Page x of y
Treatment = a single dose of 15 mg AX-158 capsules over 2 treatment periods, in the fed and fasted state.
Results obtained using an ANOVA with fixed effects of treatment, period, sequence and subject nested within sequence.


**Document Title:** SAP Template - Phase 1


#### AX-158-101 Figure 14.4.2.2

Food Effect Least Squares Geometric Mean Ratios and 90% CI of Plasma AX-158 PK Data - Part B (Food Effect)
PK Set

```
Figure Specifications

Plot type: Least squares geometric mean ratios (with 90% CI) overlaid with individual subject ratios.

By: Parameter - Cmax, AUCo-t and AUCo-inf displayed on one plot.

x axis: Parameter x axis: Label: Label each parameter including units x axis: values: 3 PK parameters (Cmax, AUCo-t, AUCo-inf)

Y axis: Least squares geometric mean ratio and 90% CI, with individual subject ratios Y axis Label: Ratio (90% CI) (%)

Y axis values: As appropriate

Legend:

15 mg AX-158 - Fed / 15 mg AX-158 - Fasted
```

Source Listing: 16.2.5.2; Produced: yyyy-mm-ddThh:mm - Page x of y
Treatment = a single dose of 15 mg AX-158 capsules over 2 treatment periods, in the fed and fasted state.
Results obtained using an ANOVA with fixed effects for fed/fasted state and subject.


**Document Title:** SAP Template - Phase 1

Document Number:TEMP-00109Previous Document Number:STATt008



# AX-158-101 Table 14.4.2.5 Summary of Statistical Analysis of Plasma AX-158 Steady State - Part C (MAD) PK Set

| | AX-158 Trough Co | ncentration ( <units>)</units> | |
|---|---|---|---|
| | Geometric I | LSMeans (95% CI) | Geometric LSMean Ratio (90% CI) |
| Treatment | Day 5 | Day 10 | Day 10/Day 5 |
| Cohort <x>:<br/>AX-158<x> mg<br/>(N=x)</x></x> | xxx<br>(xx.xx, xx.xx) | xxx<br>(xx.xx - xx.xx) | x.xx<br>(x.xx - x.xx) |
| Cohort < <i>X</i> >: AX-158< <i>X</i> > mg (N=x) | xxx<br>(xx.xx, xx.xx) | xxx<br>(xx.xx - xx.xx) | x.xx<br>(x.xx - x.xx) |

Source Listing: 16.2.5.1; Produced: yyyy-mm-ddThh:mm Page x of y

Treatment: once daily dosing of AX-158 or placebo in a <fasted/fed> state for 10 days, with the final dose administered on the morning of Day 10.

Results obtained using a mixed effects ANOVA on log-transformed data with a fixed effect of study day and a random effect of subject.


**Document Title:** SAP Template - Phase 1



#### AX-158-101 Figure 14.4.2.3

Steady State Least Squares Geometric Mean Ratios and 90% CIs of Plasma AX-158 Concentration Data - Part C (MAD)

PK Set

#### <Treatment>

#### Figure Specifications

Plot type: Least squares geometric mean ratios (with 90% CI) overlaid with individual subject ratios.

By: Treatment and comparison - Day 10/Day 5 displayed on one plot, one plot per treatment.

x axis: Parameter

x axis: Label: Comparison
x axis: values: Day 10/Day 5

Y axis: Least squares geometric mean ratio and 90% CI, with individual subject ratios

Y axis Label: Ratio (90% CI) Y axis values: As appropriate

Legend: N/a

Source Listing: 16.2.5.1; Produced: yyyy-mm-ddThh:mm - Page x of y

Treatment: once daily dosing of AX-158 or placebo in a <fasted/fed> state for 10 days, with the final dose administered on the morning of Day 10.

Results obtained using a mixed effects ANOVA on log-transformed data with a fixed effect of study day and a random effect of subject.


**Document Title:** SAP Template - Phase 1

**Document Number:** TEMP-00109 **Previous Document Number:** STATt008





 $\begin{array}{c} {\rm AX-158-101} \\ {\rm Table~14.4.2.6} \\ {\rm Summary~of~Statistical~Analysis~of~Plasma~AX-158~Accumulation~-~Part~C~(MAD)} \\ {\rm PK~Set} \end{array}$ 

| | | | Geometri<br>(95% | Geometric LSMean Ratio (90% C.I.) | |
|---|---|---|---|---|---|
| Dose Level | Parameter | n | Day 1 | Day 10 | Day 10 / Day 1 |
| Cohort <x>:</x> | C <sub>max</sub> ( <units>)</units> | Х | x.xx (x.xx, x.xx) | x.xx (x.xx, x.xx) | x.xx (x.xx, x.xx) |
| X-158 <i><x></x></i> mg<br>(N=x) | AUC <sub>0-tau</sub> ( <units>)</units> | Х | x.xx (x.xx, x.xx) | x.xx (x.xx, x.xx) | x.xx (x.xx, x.xx) |
| Cohort <x>:</x> | C <sub>max</sub> ( <units>)</units> | Х | x.xx (x.xx, x.xx) | x.xx (x.xx, x.xx) | x.xx (x.xx, x.xx) |
| AX-158 <x> mg<br/>(N=x)</x> | AUC <sub>0-tau</sub> ( <units>)</units> | Х | x.xx (x.xx, x.xx) | x.xx (x.xx, x.xx) | x.xx (x.xx, x.xx) |

Source Listing: 16.2.5.7; Produced: yyyy-mm-ddThh:mm - Page x of y

Treatment: once daily dosing of AX-158 or placebo in a < fasted/fed > state for 10 days, with the final dose administered on the morning of Day 10.

Results obtained using a mixed effects ANOVA on log-transformed data with a fixed effect of study day and a random effect of subject.


**Document Title:** SAP Template - Phase 1



AX-158-101 Figure 14.4.2.4

Accumulation Least Squares Geometric Mean Ratios and 90% CIs of Plasma AX-158 Pharmacokinetic Data - Part C (MAD)

PK Set

Day 10 / Day 1

#### Figure Specifications

Plot type: Least squares geometric mean ratios (with 90% CI) overlaid with individual subject ratios.

By: Parameter and treatment -  $C_{max}$  and  $AUC_{0-tau}$  displayed on separate plots.

x axis: Parameter

x axis: Label: AX-158 Dose (mg)
x axis: values: AX-158 dose levels

Y axis: Least squares geometric mean ratio and 90% CI, with individual subject dose-normalised values

Y axis Label: Ratio (90% CI) Y axis values: As appropriate

Source Listing: 16.2.5.7; Produced: yyyy-mm-ddThh:mm - Page x of y

Treatment: once daily dosing of AX-158 or placebo in a <fasted/fed> state for 10 days, with the final dose administered on the morning of Day 10.

Results obtained using a mixed effects ANOVA on log-transformed data with a fixed effect of study day and a random effect of subject.


**Document Title:** SAP Template - Phase 1

**Document Number:** TEMP-00109 **Previous Document Number:** STATt008



### $\begin{array}{c} {\rm AX-158-101} \\ {\rm Table~14.4.2.7} \\ {\rm Summary~of~Urine~AX-158~Concentration~Data~-~Part~C~(MAD)} \\ {\rm PK~Set} \end{array}$

| | | | | | AX | -158 Conce | ntration | n ( <units>)</units> | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | Study | | | | Geometri | .C | | | | |
| Treatment | Day | Time Interval | n | Mean | Mean | SD | %CV | Minimum | Median | Maximum |
| Cohort <x>:</x> | Х | PRE-DOSE | Х | x.xx | X.XX | x.xxx | x.x | <b>X.</b> X | x.xx | х.х |
| AX-158 <i><x></x></i> mg | | 0 н – 12 н | Х | X.XX | X.XX | x.xxx | X . X | X.X | X.XX | X.X |
| (N=x) | | 12 н – 24 н | Х | X.XX | X.XX | x.xxx | X.X | X.X | X.XX | X . X |
| | | 24 н – 48 н | X | X.XX | X.XX | X.XXX | x.x | X.X | X.XX | X.X |
| | | 48 H - 72 H | Х | X.XX | X.XX | X.XXX | X.X | X.X | X.XX | X.X |
| Cohort <x>:</x> | X | PRE-DOSE | Х | x.xx | x.xx | x.xxx | х.х | х.х | x.xx | х.х |
| AX-158 < X > mg | | 0 н – 12 н | Х | X.XX | x.xx | x.xxx | X . X | x.x | x.xx | x.x |
| (N=x) | | 12 H - 24 H | Х | x.xx | x.xx | x.xxx | X . X | x.x | X.XX | X.X |
| | | 24 H - 48 H | X | X.XX | x.xx | x.xxx | X.X | X.X | X.XX | X . X |
| | | 48 H - 72 H | Х | x.xx | x.xx | x.xxx | x.x | X . X | x.xx | x.x |

Source Listing: 16.2.5.8; Produced: yyyy-mm-ddThh:mm - Page x of y

Treatment: once daily dosing of AX-158 or placebo in a <fasted/fed> state for 10 days, with the final dose administered on the morning of Day 10.

Lower Limit of Quantitation - xx.xx < units >. BLQ values set to 0 at pre-dose and LLOQ/2 for post-dose samples. In order to capture the zero values within the calculation of the geometric mean, a value of 0.001 was added to all pre-dose values prior to log-transformation. The geometric means were then calculated and 0.001 subtracted from the estimate, i.e. geometric mean = exp (mean of log(concentration+0.001)) - 0.001.


**Document Title:** SAP Template - Phase 1



AX-158-101 Listing 16.2.1.1 Visit Dates Safety Set

Part <X> (<SAD/Food Effect/MAD - Cohort <X>: <Treatment>)

| Subject | Visit | Start Date |
|---------|---------|------------|
| XXX | xxxxxx | xxxxxx |
| | xxxxxxx | XXXXXX |
| | XXXXXXX | XXXXXX |
| | XXXXXXX | XXXXXX |
| | XXXXXXX | XXXXXX |
| XXX | XXXXXXX | XXXXXX |
| | XXXXXXX | XXXXXX |
| | XXXXXXX | XXXXXX |
| | XXXXXXX | XXXXXX |
| | XXXXXXX | XXXXXX |
| XXX | xxxxxxx | XXXXXX |
| | xxxxxxx | XXXXXX |
| | XXXXXX | XXXXXX |
| | XXXXXX | XXXXXX |
| | xxxxxx | XXXXXX |

Produced: yyyy-mm-ddThh:mm - Page x of y

Treatment: <appropriate treatment footnote for study part>

Programming Note: Cohort and treatment will not be included in the sub-header for Part B. For Part B, treatment will be included as a column within the listing.

Programming note: Listings will be repeated within an output for each part with the appropriate treatment footnote for each part.


**Document Title:** SAP Template - Phase 1



#### AX-158-101 Listing 16.2.1.2 Study Drug Administration - (1) Safety Set

Part <X> (<SAD/Food Effect/MAD - Cohort <X>: <Treatment>)

| | | Pre-Dose | | Consumed<br>Meal 30 | Fluid | Satisfy<br>Inclusion/ | Still<br>Eligible |
|---|---|---|---|---|---|---|---|
| | | Assessments | Fasted | min Prior | Withheld | Exclusion | for |
| Subject | Visit | Performed | for 10h | to Dosing | for 1h | Criteria | Dosing |
| XXX | XXXXXX | X | X | X | X | X | X |
| XXX | XXXXXX | X | Х | X | X | X | X |
| XXX | XXXXXX | X | Х | X | X | X | X |
| XXX | XXXXXX | X | X | X | X | X | X |

Produced: yyyy-mm-ddThh:mm - Page x of y

Treatment: <appropriate treatment footnote for study part>

Programming Note: Cohort and treatment will not be included in the sub-header for part B. For Part B, treatment will be included as a column within the listing.


**Document Title:** SAP Template - Phase 1



AX-158-101 Listing 16.2.1.2 Study Drug Administration - (2) Safety Set

Part <X> (<SAD/Food Effect/MAD - Cohort <X>: <Treatment>)

| | | | Dose | | Consume 240 | | | Avoided |
|---|---|---|---|---|---|---|---|---|
| | | | Admin- | | ml of water | Hand/ | Remained | Fluid |
| | | Dosing | istered | | with dose? If | Mouth | Seated | Until 1h |
| Subject | Visit | Date/Time | (mg) | Frequency | not specify. | Check | for 1h | Post-Dose |
| XXX | XXXXXX | xxxxxxTxx:xx | XXX | XXXXXX | X | X | XXX | X |
| | XXXXXX | xxxxxxTxx:xx | XXX | XXXXXX | X | X | XXX | X |

Produced: yyyy-mm-ddThh:mm - Page x of y

Treatment: <appropriate treatment footnote for study part>

Programming Note: Cohort and treatment will not be included in the sub-header for part B. For Part B, treatment will be included as a column within the listing.


**Document Title:** SAP Template - Phase 1



AX-158-101 Listing 16.2.1.3 Subject Disposition All Consented Set

Part <X> (<SAD/Food Effect/MAD - Cohort <X>: <Treatment>)

| | Informed Consent | | Screening Completion | | Study Completion/Termination | | | |
|---|---|---|---|---|---|---|---|---|
| Subject/<br>Screening<br>Number | Date/<br>Time | Version | Screening<br>Failure/<br>Non-Runner | Date<br>Randomised | Study<br>Completed | Date of<br>Completion/<br>Withdrawal | Reason for<br>Withdrawal | Comments |
| XXX | xxxxxTxx:xx | XXXX | X | XXXXXXX | X | XXXX | XXXX | XXXXXXX |
| XXX | xxxxxTxx:xx | XXXX | X | XXXXXXX | X | XXXX | XXXX | xxxxxxx |

Produced: yyyy-mm-ddThh:mm - Page x of y

Programming Note: randomised subjects should be presented before screening failures/non-runners and Subject Number will be presented for randomised subjects and Screening number for screening failures/non-runners.

For Part B, Cohort and treatment will not be included in the sub-header.


**Document Title:** SAP Template - Phase 1



AX-158-101 Listing 16.2.1.4 Additional Notes Safety Set

Part <X> (<SAD/Food Effect/MAD - Cohort <X>: <Treatment>)

| | Comment | | | |
|---|---|---|---|---|
| Subject | Number | Date | Form/Visit | Comment |
| XXX | X | XXXXXX | XXXXX-XXXXX | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | X | XXXXXX | XXXXX-XXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| | X | XXXXXX | XXXXX-XXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| | X | XXXXXX | xxxxx-xxxxx | ***************** |
| XXX | X | xxxxxx | xxxxx-xxxx | *********** |
| | Х | xxxxxx | xxxxx-xxxxx | ************* |
| | Х | XXXXXX | xxxxx-xxxxx | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| XXX | X | xxxxx | xxxxx-xxxxx | *********** |
| | X | XXXXXX | xxxxx-xxxxx | *************************************** |
| | X | XXXXXX | XXXXX-XXXXX | ****************** |
| | X | XXXXXX | xxxxx-xxxxx | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |

Produced: yyyy-mm-ddThh:mm - Page x of y

Programming Note: For Part B, cohort and treatment will not be included in the sub-header.


**Document Title:** SAP Template - Phase 1



AX-158-101 Listing 16.2.2.1 Protocol Deviations Safety Set

Part <X> (<SAD/Food Effect/MAD - Cohort <X>: <Treatment>)

| Subject | Deviation<br>Number | Date of<br>Deviation | Deviation<br>Type | Deviation | Classification |
|---|---|---|---|---|---|
| | | | * * | | |
| xxx | Х | xxxxx | xxxxxxx | xxxxxxxxxxxxxxxxxxxxxxxxxx | <major minor=""></major> |
| | X | XXXXXX | XXXXXXX | xxxxxxxxxxxxxxxxxxxxxxxxxxxx | <major minor=""></major> |
| | X | XXXXXX | XXXXXXX | xxxxxxxxxxxxxxxxxxxxxxxxxxxx | <major minor=""></major> |
| | Х | XXXXXX | XXXXXXX | xxxxxxxxxxxxxxxxxxxxxxxxxxx | <major minor=""></major> |
| XXX | Х | xxxxxx | xxxxxxxx | ****** | <major minor=""></major> |
| | X | XXXXXX | XXXXXXX | xxxxxxxxxxxxxxxxxxxxxxxxxxxx | Major/Minor> |
| | X | xxxxxx | XXXXXXX | xxxxxxxxxxxxxxxxxxxxxxxx | <major minor=""></major> |
| XXX | X | xxxxxx | xxxxxxxx | ******* | <major minor=""></major> |
| | X | XXXXXX | xxxxxxx | xxxxxxxxxxxxxxxxxxxxxxxxx | Major/Minor> |
| | X | XXXXXX | XXXXXXX | xxxxxxxxxxxxxxxxxxxxxxxxxxxx | <major minor=""></major> |
| | X | XXXXXX | XXXXXXX | xxxxxxxxxxxxxxxxxxxxxxxxxxx | <major minor=""></major> |

Produced: yyyy-mm-ddThh:mm - Page x of y

Programming Note: For Part B, cohort and treatment will not be included in the sub-header.


**Document Title:** SAP Template - Phase 1





AX-158-101 Listing 16.2.3.1 Analysis Sets All Consented Set

Part <X> (<SAD/Food Effect/MAD - Cohort <X>: <Treatment>)

| Subject/<br>Screening<br>Number | All Consented Set | Safety<br>Set | Reason for Exclusion from Safety Set | PK<br>Set | Reason for Exclusion from PK Set |
|---|---|---|---|---|---|
| XXX | Х | X | | Х | |
| XXX | X | X | | X | |
| XXX | X | X | | X | |
| XXX | X | X | | X | |
| XXX | X | X | | X | |
| XXX | X | X | | X | xxxxxxxxxxxxxxxxxxx |
| XXX | X | X | | X | |
| XXX | X | X | xxxxxxxxxxxxxxxx | Х | xxxxxxxxxxxxxxxxxxxxx |

Produced: yyyy-mm-ddThh:mm - Page x of y


**Document Title:** SAP Template - Phase 1



AX-158-101
Listing 16.2.4.1
Demographic Information
Safety Set

Part <X> (<SAD/Food Effect/MAD - Cohort <X>: <Treatment>)

| | Screening | Year of | Age | | | | Height | Weight | BMI |
|---|---|---|---|---|---|---|---|---|---|
| Subject | Number | Birth | (Yrs) | Gender | Ethnicity | Race | (m) | (kg) | (kg/m² |
| XXX | XXX | XXXXX | XXX | X | XXXXXXX | XXXXXXX | XXX | XXX | XXX |
| XXX | XXX | XXXXX | XXX | X | XXXXXX | XXXXXXX | XXX | XXX | XXX |
| XXX | XXX | XXXXX | XXX | Х | XXXXXXX | xxxxxx | XXX | XXX | XXX |

Produced: yyyy-mm-ddThh:mm - Page x of y

Programming Note: For Part B, cohort and treatment will not be included in the sub-header.


**Document Title:** SAP Template - Phase 1



AX-158-101 Listing 16.2.4.2 Substance Use History Safety Set

Part <X> (<SAD/Food Effect/MAD - Cohort <X>: <Treatment>)

| | | Average number | Date | |
|---------|-----------|----------------|---------|-----------|
| | Smoking | of cigarettes | Stopped | Smoking |
| Subject | Status | per day | Smoking | Comments |
| XXX | xxxxxxxxx | xxxxxxxxx | XXXXXX | xxxxxxxxx |
| XXX | xxxxxxxxx | xxxxxxxxx | XXXXXXX | xxxxxxxxx |
| XXX | xxxxxxxxx | xxxxxxxxx | XXXXXXX | |
| XXX | XXXXXXXXX | xxxxxxxxx | XXXXXXX | |
| XXX | xxxxxxxxx | xxxxxxxxx | XXXXXXX | |
| XXX | xxxxxxxxx | xxxxxxxxx | XXXXXXX | |
| XXX | xxxxxxxxx | xxxxxxxxx | XXXXXXX | |
| XXX | XXXXXXXXX | xxxxxxxxx | XXXXXXX | |
| XXX | XXXXXXXXX | xxxxxxxxx | XXXXXXX | xxxxxxxxx |
| XXX | xxxxxxxxx | xxxxxxxxx | XXXXXX | |
| XXX | XXXXXXXXX | xxxxxxxxx | xxxxxx | |

Produced: yyyy-mm-ddThh:mm - Page x of y

Programming Note: For Part B, cohort and treatment will not be included in the sub-header.


**Document Title:** SAP Template - Phase 1



# AX-158-101 Listing 16.2.4.3 Medical History and Concurrent Conditions Safety Set

Part <X> (<SAD/Food Effect/MAD - Cohort <X>: <Treatment>)

| | Medical | System Organ Class/ | | Date | Medication | |
|---|---|---|---|---|---|---|
| | History | Preferred Term/ | Date of | Resolved/ | Taken/Treatment | Clinically |
| Subject | Number | Reported Term | Onset | Ongoing | Currently Given? | Significant |
| ΚΧΧ | х | xxxxxxxxx/ | xxxxxxx | xxxxxxx | X | X |
| | | xxxxxxxxx/ | | | | |
| | | XXXXXXXXX | | | | |
| | X | xxxxxxxxx/ | XXXXXXX | XXXXXXX | Х | X |
| | | xxxxxxxxx/ | | | | |
| | | xxxxxxxxx | | | | |
| | X | xxxxxxxxx/ | XXXXXXX | XXXXXXX | X | X |
| | | xxxxxxxxx/ | | | | |
| | | xxxxxxxxx | | | | |

Produced: yyyy-mm-ddThh:mm - Page x of y MedDRA version <x.x>.

Programming Note: For Part B, cohort and treatment will not be included in the sub-header.


**Document Title:** SAP Template - Phase 1



AX-158-101 Listing 16.2.4.4 Virology Results Safety Set

Part <X> (<SAD/Food Effect/MAD - Cohort <X>: <Treatment>)

| | | Sample | | | | | Repeat |
|---|---|---|---|---|---|---|---|
| Subject | Visit | Date/Time | Sample ID | Source | Parameter | Result | Required |
| XXX | XXXXXX | XXXXXX | XXXXXX | <crf lab<="" td=""><td>XXXXXX</td><td>XXXXXX</td><td>X</td></crf> | XXXXXX | XXXXXX | X |
| | | Txx:xx | | Transfer> | XXXXXX | XXXXXX | X |
| | | | | | XXXXXX | XXXXXX | X |
| | | | | <crf lab<="" td=""><td>XXXXXX</td><td>XXXXXX</td><td>X</td></crf> | XXXXXX | XXXXXX | X |
| | | | | Transfer> | XXXXXX | XXXXXX | X |
| | | | | | xxxxxx | XXXXXX | Х |
| XXX | XXXXXX | xxxxxx | xxxxxx | <crf lab<="" td=""><td>xxxxx</td><td>XXXXXX</td><td>Х</td></crf> | xxxxx | XXXXXX | Х |
| | | Txx:xx | | Transfer> | XXXXXX | XXXXXX | X |
| | | | | | XXXXXX | XXXXXX | X |
| | | | | <crf lab<="" td=""><td>XXXXXX</td><td>XXXXXX</td><td>X</td></crf> | XXXXXX | XXXXXX | X |
| | | | | Transfer> | XXXXXX | XXXXXX | X |
| | | | | | XXXXXX | XXXXXX | X |

Produced: yyyy-mm-ddThh:mm - Page x of y

Programming Note: For Part B, cohort and treatment will not be included in the sub-header.


**Document Title:** SAP Template - Phase 1



AX-158-101 Listing 16.2.4.5 COVID-19 Results Safety Set

Part <X> (<SAD/Food Effect/MAD - Cohort <X>: <Treatment>)

| | | | Sample | | | | Repeat |
|---|---|---|---|---|---|---|---|
| Subject | Visit | Date/Time | ID | Source | Parameter | Result | Required |
| xxx | xxxxx | xxxxxTxx;xx | xxxxxxx | <crf <br="">Lab Transfer&gt;</crf> | xxxxxxxxx | xxxxxx | х |
| xxx | xxxxxx | xxxxxTxx:xx | xxxxxxx | <crf <br="">Lab Transfer&gt;</crf> | xxxxxxxxx | xxxxxx | Х |
| xxx | xxxxxx | xxxxxTxx:xx | xxxxxxx | <crf <br="">Lab Transfer&gt;</crf> | xxxxxxxxx | xxxxxx | Х |
| xxx | xxxxx | xxxxxTxx:xx | xxxxxxx | <crf <br="">Lab Transfer&gt;</crf> | xxxxxxxxxx | xxxxxx | Х |
| xxx | xxxxxx | xxxxxTxx:xx | xxxxxxx | <crf <br="">Lab Transfer&gt;</crf> | xxxxxxxxx | xxxxxx | х |

Produced: yyyy-mm-ddThh:mm - Page x of y

Programming Note: For Part B, cohort and treatment will not be included in the sub-header.


**Document Title:** SAP Template - Phase 1



AX-158-101 Listing 16.2.4.6 Drugs of Abuse Results Safety Set

Part <X> (<SAD/Food Effect/MAD - Cohort <X>: <Treatment>)

| | | Sample | | | | | Repeat |
|---|---|---|---|---|---|---|---|
| Subject | Visit | Date/Time | Sample ID | Source | Parameter | Result | Required |
| xxx | xxxxx | xxxxxx<br>Txx:xx | xxxxx | <crf lab<br="">Transfer&gt;</crf> | ******<br>******<br>***** | xxxxxx<br>xxxxxx<br>xxxxxx | х |
| | | | | | xxxxxx | XXXXXX | |
| | | | | <crf lab<br="">Transfer&gt;</crf> | xxxxx<br>xxxxx<br>xxxxx<br>xxxxx | xxxxx<br>xxxxx<br>xxxxx<br>xxxxx | х |

Produced: yyyy-mm-ddThh:mm - Page x of y

Programming Note: For Part B, cohort and treatment will not be included in the sub-header.


**Document Title:** SAP Template - Phase 1



# AX-158-101 Listing 16.2.4.7 Inclusion/Exclusion Criteria Failures Safety Set

Part <X> (<SAD/Food Effect/MAD - Cohort <X>: <Treatment>)

| | | Inclusion/ | Criteria | |
|---------|--------|------------|----------|--------|
| Subject | Visit | Exclusion | Number | Result |
| XXX | XXXXXX | XXXXXX | XX | xxxxx |
| XXX | XXXXXX | xxxxx | XX | XXXXXX |
| XXX | XXXXXX | XXXXXX | XX | XXXXXX |

Produced: yyyy-mm-ddThh:mm - Page x of y

Programming note: If there are no inclusion/exclusion criteria failures, display 'All subjects complied with the inclusion/exclusion criteria'.

Programming Note: For Part B, cohort and treatment will not be included in the sub-header.


**Document Title:** SAP Template - Phase 1



# AX-158-101 Listing 16.2.5.1 Plasma AX-158 Concentration Data Safety Set

Part <X> (<SAD/Food Effect/MAD - Cohort <X>: <Treatment>)

| | | | Theoretical | Actual | | AX-158 | |
|---|---|---|---|---|---|---|---|
| | | Time | Date/Time | Date/Time | Deviation | Conc. | |
| Subject | Visit | Point | of Sample | of Sample | (min) | ( <units>)</units> | Comment |
| XXX | XXXXXXXX | XX | xxxxxxTxx:xx | xxxxxxTxx:xx | XX | XXX | |
| | | XX | xxxxxxTxx:xx | xxxxxxTxx:xx | XX | XXX | |
| | | XX | xxxxxxTxx:xx | xxxxxxTxx:xx | XX | XXX | XXXXXXX |
| | | XX | xxxxxxTxx:xx | xxxxxxTxx:xx | XX | XXX | |
| | | XX | xxxxxxTxx:xx | xxxxxxTxx:xx | XX | XXX | |
| | | XX | xxxxxxTxx:xx | xxxxxxTxx:xx | XX | XXX | |
| | | XX | xxxxxxTxx:xx | xxxxxxTxx:xx | XX | XXX | XXXXXXX |
| | | XX | xxxxxxTxx:xx | xxxxxxTxx:xx | XX | XXX | |

Produced: yyyy-mm-ddThh:mm - Page x of y

Treatment: <appropriate treatment footnote for study part>

Lower Limit of Quantitation - XX.XX <units>.

Programming Note: For Part B, treatment will be included as a column within the listing.


**Document Title:** SAP Template - Phase 1



### AX-158-101 Figure 16.2.5.1 Individual Plasma AX-158 Concentration-Time Curves on a Linear Scale Safety Set

Part <X> (<SAD/Food Effect/MAD - Cohort <X>: <Treatment>

#### Figure Specifications

•

By: Treatment with all subjects on one plot, and also study day for Part C, with a separate plot for each PK profile day. For Part B, one plot per subject presenting all treatments.

x axis: Time

x axis: Label: Time (h)

x axis: values: 0 to last sampling time point (present sampling time points only)

Y axis: AX-158 concentration

Y axis Label: AX-158 Conc. ( $\langle units \rangle$ )

Y axis values: As appropriate

Legend N/A

Source Listing: 16.2.5.1; Produced: yyyy-mm-ddThh:mm - Page x of y

Treatment: <appropriate treatment footnote for study part>

Lower Limit of Quantification = xx.xx < units >. BLQ values set to zero at pre-dose and LLOQ/2 for post-dose samples. In order to capture the zero values within the calculation of the geometric mean, a value of 0.001 was added to all Day 1 pre-dose values prior to log-transformation. The geometric means were then calculated and 0.001 subtracted from the estimate, i.e. geometric mean = exp(mean of log(concentration+0.001)) - 0.001.

Programming note: Similar figures will be produced for Individual Plasma AX-158 Concentration-Time Curves on a Semi-Logarithmic Scale (Figure 16.2.5.2).


**Document Title:** SAP Template - Phase 1



## AX-158-101 Listing 16.2.5.2 Individual Derived Plasma AX-158 Pharmacokinetic Parameters Safety Set

Part <X> (<SAD/Food Effect/MAD - Cohort <X>: <Treatment>)

| Subject | Visit | Parameter | Value | Unit |
|---------|---------|-----------|-------|------|
| XXX | XXXXXXX | XXXXXXXXX | X . X | XXXX |
| | | XXXXXXXXX | X . X | XXXX |
| | | XXXXXXXXX | X . X | XXXX |
| | | XXXXXXXXX | X . X | XXXX |
| | | xxxxxxxxx | X . X | XXXX |
| | | xxxxxxxxx | X . X | XXXX |
| XXX | XXXXXXX | XXXXXXXXX | X . X | XXXX |
| | | XXXXXXXXX | X . X | XXXX |
| | | XXXXXXXXX | X . X | XXXX |
| | | xxxxxxxxx | X . X | XXXX |
| | | xxxxxxxxx | x.x * | XXXX |
| | | XXXXXXXXX | X • X | xxxx |

Produced: yyyy-mm-ddThh:mm - Page x of y

Treatment: <appropriate treatment footnote for study part>

Lower Limit of Quantification = xx.xx < units. For the purposes of PK parameter calculation, BLQ values were set to zero at pre-dose and missing for post-dose time points.

\* AUC%extrap value greater than 20%.

Programming note: A similar listing will be produced for Listing 16.2.5.9 Individual Derived Urine AX-158 Pharmacokinetic Data.


**Document Title:** SAP Template - Phase 1





AX-158-101 Listing 16.2.5.3

Raw Statistical Analysis of Plasma AX-158 Pharmacokinetic Data - Dose Proportionality
PK Set

To be populated with raw ANOVA output.

Source Listing: 16.2.5.2 Produced: yyyy-mm-ddThh:mm - Page x of y
Treatment: <appropriate treatment footnote for study part>
Results obtained using a regression analysis on log-transformed values versus log-transformed dose using the power model.

Programming Note: Similar listings will be presented for:
Listing 16.2.5.4 Raw Statistical Analysis of Plasma AX-158 Pharmacokinetic Data - Dose Independence
Listing 16.2.5.5 Raw Statistical Analysis of Plasma AX-158 Pharmacokinetic Data - Food Effect
Listing 16.2.5.6 Raw Statistical Analysis of Plasma AX-158 Pharmacokinetic Data - Steady State

Listing 16.2.5.7 Raw Statistical Analysis of Plasma AX-158 Pharmacokinetic Data - Accumulation


**Document Title:** SAP Template - Phase 1





# AX-158-101 Listing 16.2.5.8 Urine AX-158 Concentration Data Safety Set

Part C (MAD) - Cohort <X>: <Treatment>)

| Subject | Visit | Time<br>Interval | Theoretical<br>Start Date/Time<br>of Sample | Theoretical<br>End<br>Date/Time<br>of Sample | Actual<br>Start Date/Time<br>of Sample | Actual End<br>Date/Time<br>of Sample | Urine<br>Weight<br>(g) | Repeat<br>Taken |
|---|---|---|---|---|---|---|---|---|
| XXX | XXXXXXX | xx - xx | xxxxxxTxx:xx | xxxxxxTxx:xx | xxxxxxTxx:xx | xxxxxxTxx:xx | XX | XXX |
| | | xx - xx | xxxxxxTxx:xx | xxxxxxTxx:xx | xxxxxxTxx:xx | xxxxxxTxx:xx | xx | xxx |
| | | xx - xx | xxxxxxTxx:xx | xxxxxxTxx:xx | xxxxxxTxx:xx | xxxxxxTxx:xx | XX | XXX |
| | | xx - xx | xxxxxxTxx:xx | xxxxxxTxx:xx | xxxxxxTxx:xx | xxxxxxTxx:xx | XX | XXX |
| | | xx - xx | xxxxxTxx:xx | xxxxxxTxx:xx | xxxxxxTxx:xx | xxxxxxTxx:xx | XX | XXX |
| | | xx - xx | xxxxxTxx:xx | xxxxxxTxx:xx | xxxxxxTxx:xx | xxxxxxTxx:xx | XX | XXX |
| | | xx - xx | xxxxxxTxx:xx | xxxxxxTxx:xx | xxxxxxTxx:xx | xxxxxxTxx:xx | XX | XXX |
| | | xx - xx | xxxxxxTxx:xx | xxxxxxTxx:xx | xxxxxxTxx:xx | xxxxxxTxx:xx | XX | XXX |
| | | xx - xx | xxxxxTxx:xx | xxxxxxTxx:xx | xxxxxxTxx:xx | xxxxxxTxx:xx | XX | XXX |
| | | xx - xx | xxxxxxTxx:xx | xxxxxxTxx:xx | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | xxxxxxTxx:xx | XX | XXX |
| | | xx - xx | xxxxxTxx:xx | xxxxxxTxx:xx | xxxxxxTxx:xx | xxxxxxTxx:xx | XX | XXX |

Produced: yyyy-mm-ddThh:mm - Page x of y

Treatment: <appropriate treatment footnote for study part>

Lower Limit of Quantitation - XX.XX <units>.


**Document Title:** SAP Template - Phase 1



AX-158-101 Listing 16.2.7.1 Adverse Events - (1) Safety Set

Part <X> (<SAD/Food Effect/MAD - Cohort <X>: <Treatment>)

| | · | System Organ Class/ | · | · | | · | Time | · |
|---|---|---|---|---|---|---|---|---|
| | Event | Preferred Term/ | Onset Date/ | End Date/ | Date | Duration | Post Dose | |
| Subject | Number | Reported Term | Time | Time/Ongoing | Reported | (dd:hh:mm) | (dd:hh:mm) | Severity |
| .,,,,, | 37 | xxxxxxxx/ | ************* | .,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,, | ********** | 1717 • 1717 • 1717 | | ************ |
| XXX | X | | XXXXXXX | XXXXXXX | XXXXXX | xx:xx:xx | xx:xx:xx | XXXXXXX |
| | | xxxxxxxx/ | Txx:xx | Txx:xx | | | | |
| | | XXXXXXXX | | | | | | |
| XXX | Х | xxxxxxxx/ | xxxxxx | xxxxxxx | xxxxxx | xx:xx:xx | xx:xx:xx | xxxxxxx |
| | | xxxxxxxxx/ | Txx:xx | Txx:xx | | | | |
| | | xxxxxxxx | | | | | | |
| | Х | xxxxxxxx/ | XXXXXXX | XXXXXX | XXXXXX | xx:xx:xx | xx:xx:xx | XXXXXXX |
| | | xxxxxxxxx/ | Txx:xx | Txx:xx | | | | |
| | | xxxxxxxx | | | | | | |
| XXX | X | xxxxxxxx/ | xxxxxxx | xxxxxx | xxxxxx | xx:xx:xx | xx:xx:xx | XXXXXXX |
| | | xxxxxxxx/ | Txx:xx | Txx:xx | | *************************************** | | |
| | | | 177.77 | 144.44 | | | | |
| | | XXXXXXXX | | | | | | |

Produced: yyyy-mm-ddThh:mm - Page x of y

Treatment: <appropriate treatment footnote for study part>

SAE = Serious Adverse Event.

MedDRA version  $\langle x.x \rangle$ .

Programming Note: Within a study part, AEs occurring prior to first dose of study drug and placebo AEs will be pooled across cohorts and presented first.


**Document Title:** SAP Template - Phase 1



AX-158-101 Listing 16.2.7.1 Adverse Events - (2) Safety Set

Part <X> (<SAD/Food Effect/MAD - Cohort <X>: <Treatment>)

| | | System Organ Class/ | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | Event | Preferred Term/ | Relationship | | SAE | | | |
| Subject | Number | Reported Term | to Study Drug | SAE | Criteria | Action | Outcome | Comment |
| XXX | X | xxxxxxxx/ | XXXXXXX | X | XXXXXXXXXX | XXXXXX | XXXXXX | XXXXXXXX |
| | | xxxxxxxx/ | | | | | | |
| | | XXXXXXXX | | | | | | |
| XXX | X | xxxxxxxx/ | xxxxxxxx | х | xxxxxxxxxxx | xxxxxx | xxxxxx | xxxxxxxx |
| 212121 | 21 | xxxxxxxx/ | 21212121212121 | 21 | 7171717171717171717171 | 2121212121 | 2121212121 | 7111111111111111111 |
| | | XXXXXXXX | | | | | | |
| | X | xxxxxxxx/ | xxxxxxx | Х | xxxxxxxxxx | XXXXXX | XXXXXX | xxxxxxxx |
| | | xxxxxxxx/ | | | *************************************** | | *********** | *************************************** |
| | | XXXXXXXXX | | | | | | |
| | | ΛΛΛΛΛΛΛΛ | | | | | | |
| XXX | Х | xxxxxxxxx/ | xxxxxxxx | Х | XXXXXXXXXXX | XXXXXX | XXXXXX | XXXXXXXX |
| | | xxxxxxxxx/ | | | | | | |
| | | xxxxxxxx | | | | | | |

Produced: yyyy-mm-ddThh:mm - Page x of y

Treatment: <appropriate treatment footnote for study part>

SAE = Serious Adverse Event.

MedDRA version  $\langle x.x \rangle$ .

Programming Note: Within a study part, AEs occurring prior to first dose of study drug and placebo AEs will be pooled across cohorts and presented first.


**Document Title:** SAP Template - Phase 1

7.1 ---- D----

Name 1 Danes



AX-158-101 Listing 16.2.8.1 Biochemistry Data Safety Set

Part <X> (<SAD/Food Effect/MAD - Cohort <X>: <Treatment>)

| | Sample | ~ 1 | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| SIT | Sample<br>Lt Date/Time | - | Sample<br>ID | Parameter<br>(Unit) | Result | Flag | Lower | Upper | Lower | Upper | Repeat<br>Req. |
| .,,,,,,,, | .,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,, | ************ | **************** | 17 1717 | ш | 37 37 | ., .,,, | 37 37 | 77 77 | X | |
| XXXXX | | XXXXXXX | | | п | | | | | Х | |
| | TXX:XX | | | | | | | | | | |
| | | | XXXXXXX | X.XX | | X.X | X.XX | X.X | X.X | | |
| | | | XXXXXXX | X.XX | | X . X | X.XX | X.X | X.X | | |
| | | | xxxxxxx | X.XX | Lo | X.X | X.XX | X.X | X.X | | |
| | | | XXXXXXX | x.xx | H* | X.X | x.xx | X.X | X.X | | |
| | | | XXXXXXX | X.XX | | X.X | X.XX | X.X | X.X | | |
| | | | XXXXXXX | X.XX | | X.X | X.XX | X.X | X.X | | |
| | | | XXXXXXX | X.XX | | X.X | X.XX | X.X | X.X | | |
| | | | XXXXXXX | X.XX | | X.X | X.XX | X.X | X.X | | |
| | | | XXXXXXX | X.XX | L* | X.X | X.XX | X.X | X.X | | |
| | | | XXXXXXX | X.XX | | X.X | X.XX | X.X | X.X | | |
| | | | Interpretation | XXXXXX | | | | | | | |
| | xxxx | · | xxxx xxxxxxx xxxxxx | XXXX XXXXXXX XXXXXXX<br>TXX:XX XXXXXXX<br>XXXXXXXX<br>XXXXXXXX<br>XXXXXXXX | ************************************** | XXXX XXXXXXX XXXXXXX X.XX H TXX:XX XXXXXXX X.XX | XXXX XXXXXXX XXXXXXX X.XX H X.X TXX:XX XXXXXXX X.XX X.X XXXXXXXX X.XX X. | XXXX XXXXXXX XXXXXXX X.XX H X.X X.XX TXX:XX XXXXXXX X.XX X.XX XXXXXXXX X.XX X. | XXXX XXXXXXX XXXXXXX X XXX X X X X X X | XXXX XXXXXXX XXXXXXX X XXX X X X X X X | |

Produced: yyyy-mm-ddThh:mm - Page x of y

Treatment: <appropriate treatment footnote for study part>

 $H^*$  = Above alert range; H = Above normal range;  $L^*$  = Below normal range;  $L^*$  = Below alert range.

Programming Note: For Part B, treatment will be included as a column within the listing.

Programming note: Similar Listings will be produced for hematology (Listing 16.2.8.2), coagulation (Listing 16.2.8.3), urinalysis [without alert ranges] (Listing 16.2.8.4), microscopy [without alert ranges] (Listing 16.2.8.5) and other laboratory data (Listing 16.2.8.6).


**Document Title:** SAP Template - Phase 1



AX-158-101 Listing 16.2.9.1 Vital Signs Data Safety Set

Part <X> (<SAD/Food Effect/MAD - Cohort <X>: <Treatment>)

| | | | Systolic | Diastolic | Pulse | _ | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | | Blood | Blood | Rate | Oral | Respiration | | |
| | Visit/ | | Pressure | Pressure | (beats/ | Temp. | Rate | | Repeat |
| Subject | Time Point | Date/Time | (mmHg) | (mmHg) | min) | (C) | (resps/min) | Review | Taken |
| XXX | XXXXXXX | xxxxxxTxx:xx | XXX | XXX | XXX | XXX | XXX | XXXXX | X |
| | XXXXXXX | xxxxxxTxx:xx | XXX | XXX | XXX | XXX | XXX | XXXXX | X |
| | XXXXXXX | xxxxxxTxx:xx | XXX | XXX | XXX | XXX | XXX | XXXXX | X |
| | XXXXXXX | xxxxxxTxx:xx | XXX | XXX | XXX | XXX | XXX | XXXXX | |
| | XXXXXXX | xxxxxxTxx:xx | XXX | XXX | xxx H | XXX | XXX | XXXXX | X |
| | XXXXXXX | xxxxxxTxx:xx | XXX | XXX | XXX | XXX | XXX | XXXXX | X |
| | XXXXXXX | xxxxxxTxx:xx | XXX | XXX | XXX | XXX | XXX | XXXXX | X |
| | XXXXXXX | xxxxxxTxx:xx | XXX | XXX | XXX | XXX | XXX | XXXXX | |
| | XXXXXXX | xxxxxxTxx:xx | XXX | XXX | XXX | XXX | XXX | XXXXX | X |
| | XXXXXXX | xxxxxxTxx:xx | XXX | XXX | XXX | xxx L | XXX | XXXXX | X |
| | | | | | | | | | X |

Produced: yyyy-mm-ddThh:mm - Page x of y

Treatment: <appropriate treatment footnote for study part>

H = Above normal range; L = Below normal range.

Programming Note: Cohort and treatment will not be included in the sub-header for part B. For Part B, treatment will be included as a column within the listing.


**Document Title:** SAP Template - Phase 1



AX-158-101 Listing 16.2.10.1 Physical Examination Safety Set

Part <X> (<SAD/Food Effect/MAD - Cohort <X>: <Treatment>)

| Subject | Visit | Performed | Date | Time |
|---------|---------|-----------|--------|-------|
| XXX | XXXXXX | Х | XXXXXX | XX:XX |
| XXX | XXXXXX | Х | XXXXXX | xx:xx |
| XXX | XXXXXX | Х | XXXXXX | xx:xx |
| XXX | XXXXXX | Х | XXXXXX | xx:xx |
| XXX | XXXXXX | Х | XXXXXX | xx:xx |
| XXX | XXXXXX | Х | XXXXXX | XX:XX |
| XXX | XXXXXX | Х | XXXXXX | XX:XX |
| XXX | XXXXXX | Х | XXXXXX | XX:XX |
| XXX | XXXXXXX | x | XXXXXX | xx:xx |

Produced: yyyy-mm-ddThh:mm - Page x of y

Programming Note: Cohort and treatment will not be included in the sub-header for part B.


**Document Title:** SAP Template - Phase 1



AX-158-101 Listing 16.2.11.1 12-Lead ECG Data Safety Set

Part <X> (<SAD/Food Effect/MAD - Cohort <X>: <Treatment>)

| | | | | Heart | RR | PR | QRS | QT | QTcF | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Visit/ | Seq. | | Rate | Interval | Interval | Width | Interval | Interval | | Repeat |
| Subject | Time Point | No. | Date/Time | (beats/min) | (msec) | (msec) | (msec) | (msec) | (msec) | Review | Taken |
| XXX | XXXXXXXX | X | xxxxxxTxx:xx | XXX | XXX | XXX | XXX | XXX | XXX | XXXXXX | X |
| | | X | xxxxxxTxx:xx | XXX | XXX | XXX | XXX | XXX | XXX | XXXXXX | X |
| | | X | xxxxxxTxx:xx | XXX | XXX | XXX | XXX | XXX | XXX | XXXXXX | X |
| | XXXXXXXX | X | xxxxxxTxx:xx | XXX | XXX | XXX | XXX | XXX | XXX | XXXXXX | X |
| | | X | xxxxxxTxx:xx | XXX | XXX | XXX | XXX | XXX | XXX | XXXXXX | X |
| | | X | xxxxxxTxx:xx | XXX | XXX | XXX | XXX | XXX | XXX | XXXXXX | X |
| | XXXXXXX | X | xxxxxxTxx:xx | XXX | XXX | XXX | XXX | XXX | XXX | XXXXXX | X |
| | | X | xxxxxxTxx:xx | XXX | XXX | XXX | XXX | XXX | XXX | XXXXXX | X |
| | | X | xxxxxxTxx:xx | XXX | XXX | XXX | XXX | XXX | XXX | XXXXXX | X |

Produced: yyyy-mm-ddThh:mm - Page x of y

Treatment: <appropriate treatment footnote for study part>

H = Above Normal Range; L = Below Normal Range.

Programming Note: Cohort and treatment will not be included in the sub-header for part B. For Part B, treatment will be included as a column within the listing.


**Document Title:** SAP Template - Phase 1



# AX-158-101 Listing 16.2.12.1 Prior and Concomitant Medications Safety Set

Part <X> (<SAD/Food Effect/MAD - Cohort <X>: <Treatment>)

| Medication | | ATC Level 4/<br>Preferred Term/ | | Dose | | Indication/ | | Start Date | Stop Date/<br>Time/ | Admin-<br>istered |
|---|---|---|---|---|---|---|---|---|---|---|
| Subject | Number | Medication Medication | Dose | | Frequency | AE Number | Route | /Time | Ongoing | by |
| xxx | х | xxxxxxx/<br>xxxxxxxx/<br>xxxxxxxx | xxx | xx | xxxxx | xxxxxxx | xxxx | xxxxxTxx:xx | xxxxxTxx:xx | xxx |
| xxx | х | xxxxxxxx/<br>xxxxxxxx/<br>xxxxxxxx | XXX | xx | xxxxx | xxxxxxx | xxxx | xxxxxxTxx:xx | xxxxxTxx:xx | XXX |
| xxx | х | xxxxxxx/<br>xxxxxxxx/<br>xxxxxxxx | XXX | XX | xxxxxx | xxxxxxx | xxxx | xxxxxxTxx:xx | xxxxxTxx:xx | xxx |

Produced: yyyy-mm-ddThh:mm - Page x of y

Treatment: <appropriate treatment footnote for study part>

WHO DDE version <XXXXXXX>.

Programming note: Within a study part, medications taken prior to first dose of study drug, prior and ongoing medications and medications taken by placebo subjects will be pooled across cohorts and presented first.


**Document Title:** SAP Template - Phase 1





AX-158-101 Listing 16.2.14.1 PD Sampling Safety Set

Part <X> (<SAD/Food Effect/MAD - Cohort <X>: <Treatment>)

| Subject | Visit | Were the PD Blood<br>Samples taken at<br>this Visit? | Date of<br>Sample | Time of<br>Sample | Timepoint | Comment |
|---|---|---|---|---|---|---|
| XXX | xxx | xxx | xxx | xx | xxxxxx | xxxxxxx |
| xxx | XXX | xxx | xxx | XX | xxxxxx | xxxxxxx |
| XXX | XXX | xxx | xxx | XX | XXXXXX | xxxxxxx |

Produced: yyyy-mm-ddThh:mm - Page x of y

Treatment: <appropriate treatment footnote for study part>

WHO DDE version <XXXXXXX>.

Programming note: Within a study part, medications taken prior to first dose of study drug, prior and ongoing medications and medications taken by placebo subjects will be pooled across cohorts and presented first.


**Document Title:** SAP Template - Phase 1



#### 16 APPENDICES

#### 16.1 NORMAL RANGES

| Vital Sign Parameters | | |
|---|---|---|
| Parameter | Normal Range | Units |
| Pulse Rate | 40-100 | beat(s) per minute (bpm) |
| Systolic Blood pressure | 90-140 | millimetre(s) of mercury (mmHg) |
| Diastolic Blood pressure | 50-90 | millimetre(s) of mercury (mmHg) |
| Respiratory Rate | 12-18 | breath(s) per minute |
| Oral Temperature | 35.0-37.5 | degrees Celsius (°C) |

| ECG Parameters | | |
|---|---|---|
| Parameter | Normal Range | Units |
| Heart Rate (HR) | 40-100 | beat(s) per minute (bpm) |
| PR Interval | 120-220 | millisecond(s) (ms) |
| QRS Width | 70-120 | millisecond(s) (ms) |
| QT Interval | N/A | N/A |
| QTc Interval (Fridericia's Formula) | Male: 350-450 | millisecond(s) (ms) |

Version:

SAP Template - Phase 1 TEMP-00109 **Document Title:** 

**Document Number: Previous Document Number:** STATt008